Official Title: Somatic Mindfulness Training for a Healthy Workforce: Student Pilot Sample

NCT Number: NCT04122534

Document Date: 08/08/2019

## **COVER PAGE**

Official Title: Somatic Mindfulness Training for a Healthy Workforce: Student Pilot Sample

NCT Number: NCT04122534

Document Date: 08/08/2019

#### STUDY PROTOCAL

#### Includes:

- 1. Approval for Modification
- 2. Modification Request
- 3. IRB Study Protocol
- 4. Consent
- 5. Survey Items



### INSTITUTIONAL REVIEW BOARD

#### For the Protection of Human Subjects FWA 00000165

2155 Analysis Drive c/o Microbiology & Immunology Montana State University Bozeman, MT 59718 Telephone: 406-994-4706

FAX: 406-994-4303 E-mail: cherylj@montana.edu

Chair: Mark Quinn

406-994-4707 mquinn@montana.edu

Administrator:

Cheryl Johnson 406-994-4706 cherylj@montana.edu

#### MEMORANDUM \*\*\*\*\*\*\*\*\*\*\*\*

TO:

Colter Ellis, Kelly Knight, Amy Talcott, Leah Helfrich, Stephanie Zappone, Lauren

Samuel, Emma Sundeen, Madison Loft, Tristian Miller, Joshua Neu, Brenna Scott,

Andrew Z. Hassanali

FROM:

Mark Quinn Mack Jume Cy Chair, Institutional Review Board for the Protection of Human Subjects

DATE:

August 8, 2019

SUBJECT:

"Somatic Mindfulness Training for a Healthy Workforce" [CE080819]

The above proposal was reviewed by expedited review by the Institutional Review Board. This proposal is now approved. See below for follow up instructions.

Please keep track of the number of subjects who participate in the study and of any unexpected or adverse consequences of the research. If there are any adverse consequences, please report them to the committee within 3 calendar days. If there are serious adverse consequences, please suspend the research until the situation has been reviewed by the Institutional Review Board.

Any changes in the human subjects' aspects of the research should be approved by the committee before they are implemented.

It is the investigator's responsibility to inform subjects about the risks and benefits of the research. Although the subject's signing of the consent form, documents this process, you, as the investigator should be sure that the subject understands it. Please remember that subjects should receive a copy of the consent form and that you should keep a signed copy for your records.

Due to the change in the Common Rule effective January 21, 2019, you will not receive follow-up renewal forms unless your research was reviewed via full committee or is sponsored by the FDA. Enclosed is a "Project Closure Form" which we would like you to fill out and submit to our office upon completion of the research project so that we can close out the protocol. Please keep this form with your application and approval letter so that you remember to submit it at the termination of your project.

Enc.





#### **Montana State University** Institutional Review Board **Request for Minor Modifications/Amendments**

**Instructions:** E-mail completed form and all revised and/or new study documents to: cherylj@montana.edu

Note: The project's IRB-approved Research Protocol must be kept current and followed throughout the life of the project with yearly renewals. Protocols approved in the Exempt category do not require yearly renewals. All study documents are subject to review.

- 1. IRB approval number: CE080819
- 2. Project Title: Somatic Mindfulness Training for a Healthy Workforce
- Principal Investigatory Coltar Ellis and Kally E. Knight du

| Э. | Contact information (phone/e-mail): kelly.knight3@montana.edu; colter.ellis@montana.e Address (where you want approval letter sent): Department of Sociology and Anthropology, Wilson Hall 2-118 |
|---|---|
| 4. | Requesting modification/amendment to: |
| | □ Research protocol |
| | □ Consent form |
| | □ Recruitment materials |
| | □ Survey instrument, interview questions X |
| | □ Research personnel |
| | □ Other, please explain: |
| 5. | Describe the modification being requested: Note: with each requested change, provide a detailed description of where within the study documents (e.g. Research protocol, survey instrument, etc.) the changes are reflected (e.g., section, question #, etc.). |
| | We want to add the "Self-Compassion Scale" to the survey. This is a commonly used 26 |

item measure. Participants respond on a five point scale. The questions are included with this document.

| 6. I | Have these | requested | changes | been | initiated? |
|------|------------|-----------|---------|------|------------|
|------|------------|-----------|---------|------|------------|

□ No X

#### 7. How will the proposed modification(s) affect study participants? N/A

Note: Federal regulations require IRB approval prior to changing a research procedure or deviating from IRB approved documents unless it is in the best interest of or for the safety of study participants. Qualtrics Survey Software 1/16/20, 2:16 PM

## **Default Question Block**

| Almost Never 2 3 4 Almost Always I'm kind to myself when I'm experiencing suffering. Almost Never 2 3 4 Almost Always When I'm going through a very hard time, I give myself the caring and tenderness I need. Almost Never 2 3 4 Almost Always | I try to be understanding and patient towards those aspects of my personality I don't like. |
|---|---|
| 3 4 Almost Always I'm kind to myself when I'm experiencing suffering. Almost Never 2 3 4 Almost Always When I'm going through a very hard time, I give myself the caring and tenderness I need. Almost Never 2 3 4 Almost Never 2 3 4 | Almost Never |
| Almost Always | O 2 |
| Almost Always I'm kind to myself when I'm experiencing suffering. Almost Never 2 3 4 Almost Always When I'm going through a very hard time, I give myself the caring and tenderness I need. Almost Never 2 3 4 Almost Never | O 3 |
| I'm kind to myself when I'm experiencing suffering. Almost Never 2 3 4 Almost Always When I'm going through a very hard time, I give myself the caring and tenderness I need. Almost Never 2 3 4 | O 4 |
| Almost Never 2 3 4 Almost Always When I'm going through a very hard time, I give myself the caring and tenderness I need. Almost Never 2 3 4 4 | Almost Always |
| Almost Never 2 3 4 Almost Always When I'm going through a very hard time, I give myself the caring and tenderness I need. Almost Never 2 3 4 4 | |
| 2 3 4 Almost Always When I'm going through a very hard time, I give myself the caring and tenderness I need. Almost Never 2 3 4 | I'm kind to myself when I'm experiencing suffering. |
| 3 4 Almost Always When I'm going through a very hard time, I give myself the caring and tenderness I need. Almost Never 2 3 4 | ○ Almost Never |
| <ul> <li>4</li> <li>Almost Always</li> </ul> When I'm going through a very hard time, I give myself the caring and tenderness I need. <ul> <li>Almost Never</li> <li>2</li> <li>3</li> <li>4</li> </ul> | O 2 |
| <ul> <li>Almost Always</li> <li>When I'm going through a very hard time, I give myself the caring and tenderness I need.</li> <li>Almost Never</li> <li>2</li> <li>3</li> <li>4</li> </ul> | 3 |
| When I'm going through a very hard time, I give myself the caring and tenderness I need. Almost Never 2 3 4 | O 4 |
| need. Almost Never 2 3 4 | Almost Always |
| need. Almost Never 2 3 4 | |
| <ul><li>2</li><li>3</li><li>4</li></ul> | When I'm going through a very hard time, I give myself the caring and tenderness I need. |
| <ul><li>○ 3</li><li>○ 4</li></ul> | Almost Never |
| O 4 | |
| | O 3 |
| Almost Always | O 4 |
| | Almost Always |

I'm tolerant of my own flaws and inadequacies.

| ○ Almost Never |
|---|
| O 2 |
| O 3 |
| <b>4</b> |
| ◯ Almost Always |
| I try to be loving towards myself when I'm feeling emotional pain. |
| Almost Never |
| O 2 |
| O 3 |
| <b>0</b> 4 |
| O Almost Always |
| When I see aspects of myself that I don't like, I get down on myself. |
| When I see aspects of myself that I don't like, I get down on myself. Almost Never |
| O Almost Never |
| <ul><li>Almost Never</li><li>2</li></ul> |
| <ul><li>Almost Never</li><li>2</li><li>3</li></ul> |
| <ul><li>Almost Never</li><li>2</li><li>3</li><li>4</li></ul> |
| <ul><li>Almost Never</li><li>2</li><li>3</li><li>4</li></ul> |
| <ul><li>Almost Never</li><li>2</li><li>3</li><li>4</li></ul> |
| Almost Never 2 3 4 Almost Always When times are really difficult, I tend to be tough on myself. |
| Almost Never 2 3 4 Almost Always When times are really difficult, I tend to be tough on myself. Almost Never |
| Almost Never 2 3 4 Almost Always When times are really difficult, I tend to be tough on myself. Almost Never 2 |
| Almost Never 2 3 4 Almost Always When times are really difficult, I tend to be tough on myself. Almost Never |
| Almost Never 2 3 4 Almost Always When times are really difficult, I tend to be tough on myself. Almost Never 2 3 3 |

Qualtrics Survey Software

1/16/20, 2:16 PM

| I can be a bit cold-hearted towards myself when I'm experiencing suffering. — Almost Never |
|---|
| O 2 |
| O 3 |
| O 4 |
| O Almost Always |
| I'm disapproving and judgmental about my own flaws and inadequacies. |
| Almost Never |
| O 2 |
| O 3 |
| O 4 |
| Almost Always |
| I'm intolerant and impatient towards those aspects of my personality I don't like. |
| Almost Never |
| O 2 |
| O 3 |
| O 4 |
| Almost Always |
| When I'm feeling inadequate in some way, I try to remind myself that feelings of inadequacy are shared by most people. |
| Almost Never |
| O 2 |

| S Survey Software | | |
|---|---|---|
| 3 | | |
| O 4 | | |
| Almost Always | | |
| I try to see my | failings as part of the human condition. | |
| Almost Never | | |
| O 2 | | |
| O 3 | | |
| O 4 | | |
| Almost Always | | |
| When I'm down | and out, I remind myself that there are lots o<br>ke I am. | f other people in the |
| When I'm down world feeling li Almost Never 2 3 4 Almost Always | and out, I remind myself that there are lots o<br>ke I am. | f other people in the |
| world feeling li Almost Never 2 3 4 Almost Always When things ar | re going badly for me, I see the difficulties as | |
| world feeling li Almost Never 2 3 4 Almost Always When things ar everyone goes | re going badly for me, I see the difficulties as | |
| world feeling li Almost Never 2 3 4 Almost Always When things ar everyone goes Almost Never | re going badly for me, I see the difficulties as | |
| world feeling li Almost Never 2 3 4 Almost Always When things ar everyone goes Almost Never 2 | re going badly for me, I see the difficulties as | |
| world feeling li Almost Never 2 3 4 Almost Always When things ar everyone goes Almost Never | re going badly for me, I see the difficulties as | |

| When I fail at something that's important to me I tend to feel alone in my failure. |
|---|
| ○ Almost Never |
| O 2 |
| O 3 |
| O 4 |
| Almost Always |
| When I think about my inadequacies it tends to make me feel more separate and cut off from the rest of the world. |
| ○ Almost Never |
| O 2 |
| O 3 |
| O 4 |
| Almost Always |
| When I'm feeling down I tend to feel like most other people are probably happier than I am. |
| Almost Never |
| O 2 |
| ○ 3 |
| O 4 |
| Almost Always |
| When I'm really struggling I tend to feel like other people must be having an easier time of it. |
| Almost Never |
| O 2 |
| O 3 |

| <b>0</b> 4 |
|---|
| Almost Always |
| When something upsets me I try to keep my emotions in balance. |
| Almost Never |
| O 2 |
| O 3 |
| O 4 |
| ☐ Almost Always |
| When I'm feeling down I try to approach my feelings with curiosity and openness. |
| Almost Never |
| O 2 |
| O 3 |
| ○ 4 |
| Almost Always |
| When something painful happens I try to take a balanced view of the situation. |
| Almost Never |
| O 2 |
| O 3 |
| O 4 |
| ☐ Almost Always |

When I fail at something important to me I try to keep things in perspective.

Qualtrics Survey Software

1/16/20, 2:16 PM

| Almost Never |
|---|
| O 2 |
| O 3 |
| O 4 |
| O Almost Always |
| When something upsets me I get carried away with my feelings. |
| ◯ Almost Never |
| O 2 |
| O 3 |
| <b>0</b> 4 |
| O Almost Always |
| When the feeling days I took to shoop and finate or association that a sugar |
| When I'm feeling down I tend to obsess and fixate on everything that's wrong. |
| Almost Never |
| Almost Never |
| <ul><li>Almost Never</li><li>2</li></ul> |
| <ul><li>Almost Never</li><li>2</li><li>3</li></ul> |
| <ul><li>Almost Never</li><li>2</li><li>3</li><li>4</li></ul> |
| <ul><li>Almost Never</li><li>2</li><li>3</li><li>4</li></ul> |
| <ul><li>Almost Never</li><li>2</li><li>3</li><li>4</li></ul> |
| Almost Never 2 3 4 Almost Always |
| Almost Never 2 3 4 Almost Always When something painful happens I tend to blow the incident out of proportion. |
| Almost Never 2 3 4 Almost Always When something painful happens I tend to blow the incident out of proportion. Almost Never |
| Almost Never 2 3 4 Almost Always When something painful happens I tend to blow the incident out of proportion. Almost Never 2 |
| Almost Never 2 3 4 Almost Always When something painful happens I tend to blow the incident out of proportion. Almost Never 2 3 3 |

Qualtrics Survey Software

1/16/20, 2:16 PM

Qualtrics Survey Software 1/16/20, 2:16 PM

| When I fail at something important to me I become consumed by feelings of inadequacy. |
|---|
| ○ Almost Never |
| O 2 |
| ○ 3 |
| O Almost Always |

| Full | Committee | Review |
|------|------------------|--------|
| | <b>Expedited</b> | Review |

## MONTANA STATE UNIVERSITY Institutional Review Board Application for Review (revised 06/01/15)

| | ************************************** | <b>V BOARD</b><br>Ap | USE ONLY. DO NOT WRITE IN THIS AREA oproval Date: |
|---|---|---|---|
| <u>D</u> | Pate: | | |
| I. | Investigators and Associates (list all investigators person listed) | involved; | application will be filed under name of first |
| | NAME: Dr. Colter Ellis DEPT: Sociology and Anthropology COMPLETE ADDRESS: P.O. Box 172380, Bozeman, E-MAIL ADDRESS: colter.ellis@montana.edu DATE TRAINING COMPLETED:03.01.2017_ | , MT 59717 <sup>.</sup> | 2380 |
| | SIGNATURE (PI or ADVISOR): | | |
| | NAME: Dr. Kelly E. Knight DEPT: Sociology and Anthropology COMPLETE ADDRESS: P.O. Box 172380, Bozeman E-MAIL ADDRESS: kelly.knight3@montana.edu DATE TRAINING COMPLETED:03.01.2017 | n, MT 59717 | -2380 |
| | NAME: Amy Talcott DEPT: Sociology and Anthropology COMPLETE ADDRESS: P.O. Box 172380, Bozeman E-MAIL ADDRESS: amyktalcott@gmail.com DATE TRAINING COMPLETED:06.28.2018 | ı, MT 59717 | -2380 |
| | | TITLE: Ur<br>PHONE #:<br>n, MT 59717 | dergraduate Research Assistant<br>N/A<br>-2380 |
| | NAME: Stephanie Zappone DEPT: Sociology and Anthropology COMPLETE ADDRESS: P.O. Box 172380, Bozeman E-MAIL ADDRESS: stephanie.zappone@student.mor DATE TRAINING COMPLETED:12.22.2018 | PHONE #:<br>n, MT 59717<br>ntana.edu | -2380 |
| | NAME: Lauren Samuel DEPT: Sociology and Anthropology COMPLETE ADDRESS: P.O. Box 172380, Bozeman E-MAIL ADDRESS: laurenlizsamuel@gmail.com DATE TRAINING COMPLETED:1.19.2019_ | :# PHONE<br>1, MT 59717 | -2380 |
| | NAME: Emma Sundeen DEPT: Sociology and Anthropology COMPLETE ADDRESS: P.O. Box 172380, Bozeman E-MAIL ADDRESS: emma.sundeen@gmail.com DATE TRAINING COMPLETED: 2.7.2019 | PHONE #:<br>n, MT 59717 | |

| C<br>E | NAME: Madison Loft DEPT: Sociology and Anthropology COMPLETE ADDRESS: P.O. Box 172380, Bozeman E-MAIL ADDRESS: themadisonloft@gmail.com DATE TRAINING COMPLETED:1.8.2018 | PHONE #:<br>, MT 59717 | |
|---|---|---|---|
| C<br>E | DEPT: Sociology and Anthropology<br>COMPLETE ADDRESS: P.O. Box 172380, Bozeman<br>E-MAIL ADDRESS: tmiller1296@gmail.com | PHONE #:<br>, MT 59717 | 7-2380 |
| Ľ | DATE TRAINING COMPLETED:6.12.2019_ | | [Required training: CITI Training; see website for link] |
| C | JAME: Joshua Neu TITLE: DEPT: Sociology and Anthropology COMPLETE ADDRESS: P.O. Box 172380, Bozeman E-MAIL ADDRESS: joshuaneu2010@gmail.com | Undergrad<br>PHONE #<br>, MT 59717 | luate Research Assistant<br>: N/A<br>7-2380 |
| C | DATE TRAINING COMPLETED:3.13.2019_ | | [Required training: CITI Training; see website for link] |
| C | IAME: Brenna Scott TITLE: DEPT: Sociology and Anthropology COMPLETE ADDRESS: P.O. Box 172380, Bozeman E-MAIL ADDRESS: bren0316@gmail.com | , MT 59717 | 7-2380 |
| | | | [Required training: CITI Training; see website for link] |
| C | AME: Andrew Z. Hassanali TITLE: DEPT: Sociology and Anthropology COMPLETE ADDRESS: P.O. Box 172380, Bozeman E-MAIL ADDRESS: andrew.hassanali@icloud.com | Research<br>PHONE #:<br>, MT 59717 | Assistant<br>: N/A<br>7-2380 |
| | OATE TRAINING COMPLETED:6.20.2019_ | | [Required training: CITI Training; see website for link] |
| (r | repeat for additional investigators if needed; or delete | xtra if not r | necessary) |
| resp | | alue or great | ir family members have consulting agreements, managemen<br>er than 5% total equity) in the sponsor, subcontractor or in<br>NO |
| If yo | ou answered <u>Yes,</u> you will need to contact Kellie Peterson, | Assistant Le | gal Counsel-JD at 406-994-3480. |
| II. | Title of Proposal: Somatic Mindfulness Training for | a Healthy | Workforce. |
| III. | Beginning Date for Use of Human Subjects: August | 15, 2019 | |
| IV. | Type of Grant and/or Project (if applicable) Research Grant: X Contract: Training Grant: Classroom Experiments/Projects: Thesis Project: Other (Specify): | | |
| V. | Name of Funding Agency to which Proposal is | Being Sul | omitted (if applicable): |

We have submitted a proposal to MSU's Center for American Indian and Rural Health Equity (CAIRHE) which is funded by the National Institutes of Health.

#### VI. Signatures

Submitted by Investigator

Typed Name: Colter Ellis, Joint-PI

Signature:

Date: 7/24/19

Faculty sponsor (for student)

Kely & hit

Typed Name: Kelly Knight, Joint-PI

Signature:

Date: 7/24/19

VII. Summary of Activity. Provide answers to each section and add space as needed. Do not refer to an accompanying grant or contract proposal.

A. RATIONALE AND PURPOSE OF RESEARCH. (What question is being asked?)

Victims of sexual assault, intimate partner violence, child neglect, and other forms of abuse depend on service providers to help them find safety, access resources, and seek justice. This work is critically important to survivors but often has negative consequences for individuals who assist them. As a result, a burgeoning body of literature has tried to document the emotional strain of this work (see Elwood, Mott, Lohr, & Galovski, 2011; Molnar et al., 2017; Sabin-Farrell & Turpin, 2003, for reviews). We define "secondary trauma" as the result of repeated empathetic engagement with traumatized populations. When workers burnout, it increases operating costs for organizations and decreases the quality of services provided (Powell and York 1992; Ullman and Townsend 2007). The scholarship, however, has yet to fully theorize the occupational hazards of victim service provision and there are few theoretically and empirically driven solutions (Bercier & Maynard, 2015). This research seeks to develop, pilot, and evaluate an intervention response that will help mitigate the negative impacts of secondary trauma.

B. RESEARCH PROCEDURES INVOLVED. Provide a short description of sequence and methods of procedures that will be performed with human subjects. Include details of painful or uncomfortable procedures, frequency of procedures, time involved, names of psychological tests, questionnaires, restrictions on usual life patterns, and follow up procedures. If you are planning on posting flyers, posters, etc. anywhere on Campus, you must check with the building managers and/or departments located in MSU buildings and obtain their approval prior to the posting.

This proposed research will develop and pilot a somatically-oriented mindfulness curriculum designed to reduce the symptoms of occupational-based secondary trauma (ST) among victim service providers working in Montana. The content of the curriculum will be based on our previously published text *Secondary Trauma in the Workplace: Tools for Awareness, Self-Care, and Organizational Response in Montana* we wrote with a group of seven local victim service providers. The curriculum for this intervention, however, will be expanded to more fully include mindfulness meditation and somatic-based trauma resolution techniques.

The intervention curriculum will be developed and tested with three cohorts.

For the **first cohort**, Drs. Knight and Ellis will pilot the curriculum in an undergraduate course in the Fall of 2019 (n= approximately 15 students). Dr. Knight will be the instructor of record. The content and effectiveness of the course will be evaluated using a survey. The complete survey and consent form are included in this application. There will be three waves of survey data collected. For the first two waves, students will be asked to complete the survey during the semester (wave one, during the first few weeks of class and wave two during the final few weeks of class). Students can choose not to complete the survey with no penalty. If at least 85%

of the students in each class participate in data collection waves one and two, all students will be eligible for some form of extra credit and/or participation in some kind of celebration (such as pizza on the last day of class). All students will be eligible, even if they themselves did not participate. A third wave may also be collected approximately one month after the course. Participation for this final wave of data collection will be incentivized by a \$20 e-gift card. Students' participation will be strictly optional.

The **second cohort** will occur in the Spring of 2020. Drs. Knight and Ellis will, again, pilot the intervention in an undergraduate course (n=35). Dr. Ellis will be the instructor of record. Again, the content and effectiveness of the course will be evaluated using a survey. Just as before, there will be three waves of survey data collected. For the first two waves, students will be asked to complete the survey during the semester (wave one, during the first few weeks of class and wave two during the final few weeks of class). Students can choose not to complete the survey with no penalty. If at least 85% of the students in each class participate in data collection waves one and two, all students will be eligible for some form of extra credit and/or participation in some kind of celebration (such as pizza on the last day of class). All students will be eligible, even if they themselves did not participate. A third wave may also be collected approximately one month after the course. Participation for this final wave of data collection will be incentivized by a \$20 e-gift card. Students' participation will be strictly optional.

After preliminary analysis of the first two student-cohorts is complete, the content will be modified as necessary and the curriculum will be piloted with a **third cohort**. This cohort will comprise of a small sample of local victim service providers. By victim service providers we mean any profession or volunteer position that involves interacting with victims of crime. These positions include, but are not limited to, law enforcement, attorneys, child protective services, healthcare providers, victim advocates, and religious clergy. Our goal is to have a small sample of 5-20 victim service providers willing to meet once a week for 15 weeks. During these meetings, we will implement our curriculum. The intervention will be evaluated by asking participants to complete the survey three times (before the training begins, at the end of the training, and then a third time one to three months post-training). Participation in this program will be incentivized with three \$20 e-gift cards, sent after each of the three surveys.

All the measures included in the survey are well established in the literature. Table 1 provides a list of measures included.

Table 1: Names of Survey Questionnaires

| Measurement Name | Abbreviation | Number of Items |
|---|---|---|
| Basic Demographics, VSP* | BD | 11 |
| Basic Demographics, Student* | BDS | 12 |
| Work Demographics* | WD | 7 |
| Maslach Burnout Inventory – General Version* | MBI-G | 16 |
| Maslach Burnout Inventory – General Student Version* | MBI-GS | 17 |
| Maslach Burnout Inventory – Student Version* | MBI-S | 16 |
| Secondary Traumatic Stress Scale | STSS | 18 |
| The PTSD Checklist for DSM-5 | PCL-5 | 20 |
| Body Mass Index | BMI | 2 |
| Health Related Quality of Life | HRQoL | 4 |
| Autoimmune Diagnosis | AD | 1 |
| Patient Health Questionnaire – Somatic Symptom Severity | PHQ-15 | 15 |
| AUDIT Alcohol Questionnaire | AUDIT | 10 |
| Tobacco, Alcohol, Prescription and Other Substance Use Tool | TAPS | 4 |
| Jenkins Sleep Scale | JSS | 4 |
| Generalized Anxiety Disorder | GAD-7 | 7 |
| Patient Health Questionnaire – Depression | PHQ-8 | 8 |
| Mental Health Specialist | MHS | 1 |
| Interpersonal Reactivity Index | IRI | 28 |
| BRFSS Adverse Childhood Experience (ACE) Module | BRFSS ACE | 11 |
| Brief Resilience Scale | BRS | 6 |
| Experiences in Close Relationships - Relationship Structures | ECR-RS | 9 |
| Multidimensional Assessment of Interoceptive Awareness | MAIA | 37 |
| Five Facets of Mindfulness Questionnaire | FFMQ | 20 |
| Trauma Exposure and Training | TE | 4 |
| Feedback | FE | 2 |

Note: \*All items may not actually appear in each survey.

C. DECEPTION - If any deception (withholding of complete information) is required for the validity of this activity, explain why this is necessary and attach debriefing statement.

No deceptive practices will be used.

#### D. SUBJECTS

1. Approximate number and ages

How Many Subjects: 65

Age Range of Subjects: 18 years and older

How Many Normal/Control: n/a

Age Range of Normal/Control: 18 years and older

2. Criteria for selection:

Study participants must be either students at MSU or working or volunteering in a victim service profession or organization. All participants must be 18 years or older.

3. Criteria for exclusion:

For the first two cohorts, those who are not undergraduate students at Montana State University will be excluded from data collection. For the third cohort, study participants not working or volunteering in a victim service profession or organization will be excluded from data collection. Anyone who is not 18 years or older will be excluded from all parts of the study.

4. Source of Subjects (including patients):

For cohorts one and two, study participants will be recruited in the classroom. Both Drs. Ellis and Knight are popular teachers who attract students interested in issues of trauma and mindfulness. For cohort 3, community contacts, victim service organizations, and community advisory board members will help with recruitment.

5. Who will approach subjects and how? Explain steps taken to avoid coercion.

Students who choose to enroll in the class will be required to read and work with the content of the course, however, they will not be required to participate in the evaluation survey. We will emphasize in the syllabus and verbally in class, that participation, or nonparticipation, in the survey is absolutely optional and will not count towards their grade in anyway. Victim service providers will be free not to participate and can end participation at any time.

6. Will subjects receive payments, service without charge, or extra course credit? **X Yes** or No (If yes, what amount and how? Are there other ways to receive similar benefits?)

For the first two cohorts, if at least 85% of the students in each class participate in data collection waves one and two, all students will be eligible for some form of extra credit and/or participation in some kind of celebration (such as pizza on the last day of class). All students will be eligible, even if they themselves did not participate. Students who participate in data collection wave three (approximately1 month after class has ended) will receive a \$20 e-gift card. Victim service providers who participate in cohort three will be eligible for MSU continuing education credits and \$20 e-gift cards for each survey.

7. Location(s) where procedures will be carried out.

Cohorts one and two will be carried out in a classroom on campus. Cohort three will be held at a time and place convenient for all the participating victim service providers.

#### E. RISKS AND BENEFITS (ADVERSE EFFECTS)

1. Describe nature and amount of risk and/or adverse effects (including side effects), substantial stress, discomfort, or invasion of privacy involved.

Some of the questions on the survey will ask about personal and potentially emotional topics. While these questions may cause some discomfort, a list of resources will be provided should participants feel they need to seek help.

While it is not the focus of the study, the survey will ask about alcohol and other drug use. We ask these questions because respondents may be using substances to cope with secondary trauma. To protect participants, identifying information will be separated from their responses and all information will be deidentified when presented or published.

2. Will this study preclude standard procedures (e.g., medical or psychological care, school attendance, etc.)? If yes, explain.

No.

3. Describe the expected benefits for individual subjects and/or society.

Survey data will document the prevalence of ST and its correlates. If successful, the intervention will be a useful tool for improving the work lives and psychological health of victim service providers.

#### F. ADVERSE EFFECTS

1. How will possible adverse effects be handled?

No adverse effects are expected. If participants become upset during the survey, a list of resources is provided in the consent form.

By investigator(s):

NA

Referred by investigator(s) to appropriate care:

N/A

Other (explain):

N/A

- 2. Are facilities/equipment adequate to handle possible adverse effects? **X Yes** or No (If no, explain.)
- 2. Describe arrangements for financial responsibility for any possible adverse effects.

None. In our view, there is no reasonable concern that a participant would experience any adverse effects.

MSU compensation (explain): NA Sponsoring agency insurance: NA Subject is responsible: NA

Other (explain): NA

#### G. CONFIDENTIALITY OF RESEARCH DATA

1. Will data be coded? X Yes or No.

- 2. Will master code be kept separate from data? X Yes or No
- 3. Will any other agency have access to identifiable data? Yes or **X No** (If yes, explain.)

Workplaces will not have access to providers' data.

4. How will documents, data be stored and protected? Locked file:

Yes, all physical files will be locked in a cabinet and in a locked office on campus.

Computer with restricted password:

Yes, all de-identified digital files will be kept on password-protected computers or stored on a secured server.

Other (explain): N/A

- VIII. Checklist to be completed by Investigator(s)
  - A. Will any group, agency, or organization be involved? Yes or **X No** (If yes, please confirm that appropriate permissions have been obtained.)
  - B. Will materials with potential radiation risk be used (e.g. x-rays, radioisotopes)? Yes or **X No** 
    - 1. Status of annual review by MSU Radiation Sources Committee (RSC). Pending or Approved (If approved, attach one copy of approval notice.)
    - 2. Title of application submitted to MSU RSC (if different).
  - C. Will human blood be utilized in your proposal? Yes or **X No** (If yes, please answer the following)
    - Will blood be drawn? Yes or X No
       (If yes, who will draw the blood and how is the individual qualified to draw blood?
       What procedure will be utilized?)
    - 2. Will the blood be tested for HIV? Yes or X No.
    - 3. What disposition will be made of unused blood?
    - 4. Has the MSU Occupational Health Officer been contacted? Yes or X No
  - D. Will non-investigational drugs or other substances be used for purposes of the research? Yes or **X No**

Name:
Dose:
Source:
How Administered:
Side effects:

| Ε. | Will any investigational new drug or other investigational substance be used? Yes or <b>X No</b> |
|---|---|
| | [If yes, provide information requested below and one copy of: 1) available toxicity data; 2) reports of animal studies; 3) |
| | description of studies done in humans; 4) concise review of the literature prepared by the investigator(s); and 5) the drug |
| | protocol.] |

Name: Dose:

Source:

How Administered:

IND Number:

Phase of Testing:

- F. Will an investigational device be used? Yes or **X No** (If yes, provide name, source description of purpose, how used, and status with the U.S. Food and Drug Administration FDA). Include a statement as to whether or not device poses a significant risk. Attach any relevant material.)
- G. Will academic records be used? Yes or X No
- H. Will this research involve the use of:

Medical, psychiatric and/or psychological records Yes or X No

Health insurance records Yes or X No

Any other records containing information regarding personal health and illness Yes or X No

If you answered "Yes" to any of the items under "H.", you must complete the **HIPAA worksheet**.

- I. Will audio-visual or tape recordings or photographs be made? Yes or X No
- J. Will written consent form(s) be used? (**X Yes** or No. If no, explain.) (Please use accepted format from our website. Be sure to indicate that participation is voluntary. Provide a stand-alone copy; do

#### List of Attachments

There are two versions of our evaluation survey, one for MSU Students and another of victim service providers. Full copies of both of these surveys are included as electronic attachments in this application.

- 02 MBTHW Student Survey Final 07.24.2019
- 03 MBTHW VSP Survey Final 07.24.2019

#### Consent, Montana VSPs

#### Hello!

This survey has been developed by Associate Professors from Montana State University to study secondary trauma.

The purpose of this study is to better understand the personal histories and experiences of victim service providers, or those considering becoming victim service providers, in Montana.

Any insights you could offer are greatly appreciated!

Before we begin, however, we need to review this consent form. This insures that your rights are protected as a participant this study.

Kelly Knight, PhD, and Colter Ellis, PhD Principal Investigators

#### Questions? We have answers:

#### Why am I being asked to participate?

You are being asked to participate in a research study because of your involvement in, or knowledge of, services in your area.

#### Why is this research being done?

This survey is being conducted to evaluate a new educational program. The program is intended to teach people strategies for managing the negative consequences of secondary trauma. Your participation will help us better understand how the personal histories and experiences of service providers impact their work and mental and physical health.

#### How long will it take me to participate?

This survey should take approximately 30-45 minutes to complete.

#### Will I be compensated for participation?

You will receive a \$20 eGift Card when you have completed the surveys.

Please allow one week for us to email you the eGift Card. Thanks for your patience with us!

#### What will I be asked to do?

Your participation in this research is voluntary and completely your choice. If you agree, you

will be asked to answer a number of questions about your personal history, your work, your physical and psychological health, and your resilience. You will also be asked to complete some basic demographic questions. You can choose to not answer any questions you do not want to answer. Also, you can stop at any time with no consequences.

#### Are there any benefits to me if I participate in this study?

This study is of no direct benefit to you. However, the information gained will inform the development of a data-driven intervention to lessen the impacts of secondary trauma on service providers.

#### Will my information be kept private?

Everything you tell us will be kept confidential. Your answers will be separated from your name and contact information (which we need to give you your eGift Card).

All data collected will be secured on a password-protected and firewalled computer in a locked office on Montana State University's campus or stored on a secure server. No one but the official research staff will have access to the information. Your results will be grouped with other participants' data when results of this study are published. Your identity will remain anonymous.

An exception to confidentiality is the indication of imminent harm to yourself or others.

#### Who should I contact if I have questions?

You can contact the principal investigators about the study: Kelly E. Knight, PhD, (406) 994-7224, kelly.knight3@montana.edu, or Colter Ellis, PhD, (406) 994-4219, colter.ellis@montana.edu. They can also be reached by mail at: Montana State University, Department of Sociology and Anthropology, PO Box 172380, Bozeman, MT, 59817.

In addition, you can contact MSU's institutional review board chairperson: Mark Quinn, PhD, (406) 994-4747, mquinn@montana.edu. He can also be reached by mail at Montana State University, IRB, PO BOX 173610, Bozeman, MT, 59817.

#### What happens if I change my mind?

Participation is strictly voluntary and you can stop at any time. Participation or non-participation will not affect your current or future relationship with Montana State University.

#### Are there any risks to me if I participate in this study?

We do not foresee any significant physical or psychological risks as a result of your participation. However, some of the questions are personal and may provoke an emotional response. Below is a list of resources should you be worried or need support after the survey.

#### **Resource List:**

1. Montana Suicide Prevention Lifeline: (800) 273-8255

- 2. MSU Voice Center: (406) 994-7069
- 3. Counseling and Psychological Services, MSU: (406) 994-4531
- 4. HELP Center Crisis and Referral Line: (406) 586-3333 or just dial 2-1-1
- 5. Haven Domestic Violence Program: (406) 586-4111
- 6. Alcohol and Drug Services of Gallatin County: (406) 586-5493
- 7. Bozeman Health Deaconess Hospital: (406) 414-5000
- 8. Bridger Care, Reproductive & Sexual Healthcare & Education: (406) 587-0681
- 9. Child and Family Services: (866) 820-5437
- 10. Gallatin Valley Mental Health Center: (406) 556-6500

#### **ELECTRONIC CONSENT:**

- You voluntarily agree to participate.
- You are 18 years of age or older.
- Agree

#### **Demographics**

What is your age?

What is your sex/gender?

Female

Male

Other

| What is the highest level of education that you have completed? |
|-----------------------------------------------------------------|
| O Did not complete high school |
| High school or equivalent |
| Some college or post high school training |
| Associate's or 2-year degree |
| Bachelor's degree |
| ○ Graduate/professional degree |
| What race do you consider yourself? Check all that apply. |
| American Indian |
| ☐ Alaskan Native |
| ☐ Asian |
| Black or African American |
| ☐ Hispanic or Latino |
| ☐ Native Hawaiian, Other Pacific Islander |
| ☐ White |
| Other |
| What is your current marital status? |
| ○ Married |
| Living with partner (but not married) |
| O Divorced/separated |
| ◯ Single |
| ○ Widowed |
| Other |

Which category best describes **your** current income from all sources before taxes?

| Oo you own or rent your home? Own Rent How long have you lived in this area? | Survey Software | | 8/6/19 |
|---|---|---|---|
| oo you own or rent your home? Own Rent No you long have you lived in this area? Oo you have a documented disability? Check all that apply. No ADHD/ADD Learning disability Psychological disability Traumatic brain injury Other Oo you consider yourself to be a veteran? | | | |
| oo you own or rent your home? Own Rent No you long have you lived in this area? Oo you have a documented disability? Check all that apply. No ADHD/ADD Learning disability Psychological disability Traumatic brain injury Other Oo you consider yourself to be a veteran? | | | |
| oo you own or rent your home? Own Rent No you long have you lived in this area? Oo you have a documented disability? Check all that apply. No ADHD/ADD Learning disability Psychological disability Traumatic brain injury Other Oo you consider yourself to be a veteran? | Which categor | best describes your total <b>2018 household</b> income from all sources before | |
| Oo you own or rent your home? Own Rent Oo you long have you lived in this area? Oo you have a documented disability? Check all that apply. No ADHD/ADD Learning disability Peychological disability Traumatic brain injury Other Oo you consider yourself to be a veteran? | taxes? | | |
| Own Rent How long have you lived in this area? O you have a documented disability? Check all that apply. No ADHD/ADD Learning disability Psychological disability Traumatic brain injury Other Oo you consider yourself to be a veteran? | | | |
| Own Rent How long have you lived in this area? O you have a documented disability? Check all that apply. No ADHD/ADD Learning disability Psychological disability Traumatic brain injury Other Oo you consider yourself to be a veteran? | Do vou own or | rent vour home? | |
| Rent How long have you lived in this area? Do you have a documented disability? Check all that apply. No ADHD/ADD Learning disability Psychological disability Traumatic brain injury Other Do you consider yourself to be a veteran? | | rent your nome? | |
| How long have you lived in this area? Do you have a documented disability? Check all that apply. No ADHD/ADD Learning disability Psychological disability Traumatic brain injury Other Do you consider yourself to be a veteran? | | | |
| Oo you have a documented disability? Check all that apply. No ADHD/ADD Learning disability Psychological disability Traumatic brain injury Of Other Oo you consider yourself to be a veteran? | Rent | | |
| Oo you have a documented disability? Check all that apply. No ADHD/ADD Learning disability Psychological disability Traumatic brain injury Of Other Oo you consider yourself to be a veteran? | | | |
| Oo you have a documented disability? Check all that apply. No ADHD/ADD Learning disability Psychological disability Traumatic brain injury Other | How long have | you lived in this area? | |
| No ADHD/ADD Learning disability Psychological disability Traumatic brain injury Other Oo you consider yourself to be a veteran? | | | |
| No ADHD/ADD Learning disability Psychological disability Traumatic brain injury Other Oo you consider yourself to be a veteran? | | | |
| ADHD/ADD Learning disability Psychological disability Traumatic brain injury Other Oo you consider yourself to be a veteran? | Do you have a | documented disability? Check all that apply. | |
| Learning disability Psychological disability Traumatic brain injury Other Oo you consider yourself to be a veteran? | No | | |
| Psychological disability Traumatic brain injury Other Oo you consider yourself to be a veteran? | ADHD/ADD | | |
| Other Oo you consider yourself to be a veteran? | Learning disability | | |
| Other Oo you consider yourself to be a veteran? | Psychological disa | ility | |
| Oo you consider yourself to be a veteran? | Traumatic brain inj | ry | |
| | Other | | |
| ) No | Do you conside | r yourself to be a veteran? | |
| | ) No | | |

## Work Demographics, VSPs

| Using these U.S. Department of Labor categories, which best describes your occupation? |
|---|
| Community and social services occupations (e.g., social workers, counselors, therapists, clergy) |
| Education, training, and library occupations (e.g., teachers, librarians) |
| Healthcare practitioners and technical occupations (e.g., physicians, nurses, paramedics) |
| Healthcare support occupations (e.g., home health aides, massage therapists) |
| Legal occupations (e.g., lawyers, judges, paralegals) |
| Protective service occupations (e.g., police officers, fire fighters, correctional officers) |
| Other |
| Please select other occupational category. |
| Architecture and Engineering Occupations |
| Arts, Design, Entertainment, Sports, and Media Occupations |
| Building and Grounds Cleaning and Maintenance Occupations |
| Business and Financial Operations Occupations |
| Computer and Mathematical Occupations |
| Construction and Extraction Occupations |
| Farming, Fishing, and Forestry Occupations |
| Food Preparation and Serving Related Occupations |
| ☐ Installation, Maintenance, and Repair Occupations |
| Life, Physical, and Social Science Occupations |
| Management Occupations |
| Office and Administrative Support Occupations |
| Personal Care and Service Occupations |
| O Production Occupations |
| Sales and Related Occupations |
| Transportation and Material Moving Occupations |
| Other |

How long have you worked in your general profession?

| Overall, how long have you worked at your current organization? |
|---|
| What is your current job title? |
| How long have you worked in your present position? |
| Is your position considered: (Please select one) Front-line staff Supervisor |
| Management (First-level) Management (Intermediate) Management (Senior) Other |
| MBI (Burnout) On this page are statements of job-related feelings. Please read each statement carefully and |

Qualtrics Survey Software

8/6/19, 7:38 PM

| | Never | A few<br>times a<br>year or<br>less | Once a<br>month or<br>less | A few times<br>a month | Once a week | A few<br>times a<br>week | Every day |
|---|---|---|---|---|---|---|---|
| I feel emotionally drained from my work. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| I feel used up at the end of the workday. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I feel tired when I get up in the morning and have to face another day on the job. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Working all day is really a strain for me. | 0 | 0 | 0 | $\circ$ | $\circ$ | 0 | |
| I can effectively solve the problems that arise in my work. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I feel burned out from my work. | 0 | 0 | 0 | 0 | $\circ$ | 0 | 0 |
| I feel I am making an effective contribution to what this organization does. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I have become less interested in my work since I started this job. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

Copyright ©1996 Wilmar B. Schaufeli, Michael P. Leiter, Christina Maslach & Susan E. Jackson. All rights reserved in all media. Published by Mind Garden, Inc., www.mindgarden.com

On this page are statements of job-related feelings. Please read each statement carefully and decide if you ever feel this way about your job.

| | Never | A few times a<br>year or less | Once a month or less | A few times a month | Once a week | A few times a week | Every day |
|---|---|---|---|---|---|---|---|
| I have become less enthusiastic about my work. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| In my opinion, I am good at my job. | $\circ$ | $\circ$ | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I feel exhilarated when I accomplish something at work. | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I have accomplished many worthwhile things in this job. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | 0 |
| I just want to do my job and not be bothered. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | 0 |
| I have become more cynical about whether my work contributes anything. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| I doubt the significance of my work. | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| At my work, I feel confident that I am effective at getting things done. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

Copyright ©1996 Wilmar B. Schaufeli, Michael P. Leiter, Christina Maslach & Susan E. Jackson. All rights reserved in all media. Published by Mind Garden, Inc., www.mindgarden.com

#### STSS (Secondary Traumatic Stress Scale)

The following is a list of statements made by persons who have been impacted by their work with traumatized clients (or other potentially traumatized populations, e.g., patients, students, customers, or anyone to whom you provide services).

In the past seven days, how frequently was the statement true for you:

| | Never | Rarely | Occasionally | Often | Very often |
|---|---|---|---|---|---|
| I felt emotionally numb. | 0 | 0 | 0 | 0 | 0 |
| My heart started pounding when I thought about my work with clients. | 0 | $\circ$ | 0 | $\circ$ | 0 |
| It seemed as if I was reliving the trauma(s) experienced by my client(s). | 0 | $\circ$ | 0 | $\circ$ | 0 |
| I had trouble sleeping. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| I felt discouraged about the future. | 0 | $\circ$ | 0 | $\circ$ | |
| Reminders of my work with clients upset me. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| I had little interest in being around others. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| I felt jumpy. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| I was less active than usual. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| I thought about my work with clients when I didn't intend to. | 0 | 0 | 0 | $\circ$ | |
| I had trouble concentrating. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| I avoided people, places, or things that reminded me of my work with clients. | 0 | $\circ$ | 0 | $\circ$ | 0 |
| I had disturbing dreams about my work with clients. | 0 | 0 | 0 | $\circ$ | |
| I wanted to avoid working with some clients. | 0 | 0 | 0 | $\circ$ | |
| I was easily annoyed. | 0 | 0 | 0 | $\circ$ | |
| I expected something bad to happen. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| I noticed gaps in my memory about client sessions. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Please select 'Very often' for this response. | 0 | 0 | 0 | $\circ$ | 0 |

#### PCL-5 (PTSD)

Below is a list of problems that people sometimes have in response to a very stressful experience. Please read each problem carefully and then indicate how much you have been bothered by that problem in the past month.

| in the <b>past month</b> , now much were you bothere | а ву: | | | | |
|---|---|---|---|---|---|
| | Not at all | A little bit | Moderately | Quite a bit | Extremely |
| Repeated, disturbing, and unwanted memories of the stressful experience? | 0 | 0 | 0 | 0 | 0 |
| Repeated, disturbing dreams of the stressful experience? | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Suddenly feeling or acting as if the stressful experience were actually happening again (as if you were actually back there reliving it)? | 0 | $\circ$ | $\circ$ | 0 | $\circ$ |
| Feeling very upset when something reminded you of the stressful experience? | 0 | $\circ$ | $\circ$ | 0 | $\circ$ |
| Having strong physical reactions when something reminded you of the stressful experience (for example, heart pounding, trouble breathing, sweating)? | 0 | 0 | 0 | 0 | 0 |
| Avoiding memories, thoughts, or feelings related to the stressful experience? | 0 | $\circ$ | $\circ$ | 0 | $\circ$ |
| Avoiding external reminders of the stressful experience (for example, people, places, conversations, activities, objects, or situations)? | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Trouble remembering important parts of the stressful experience? | 0 | | 0 | 0 | 0 |
| Having strong negative beliefs about yourself, other people, or the world (for example, having thoughts such as: I am bad, there is something seriously wrong with me, no one can be trusted, the world is completely dangerous)? | 0 | 0 | 0 | 0 | 0 |
| Blaming yourself or someone else for the stressful experience or what happened after it? | 0 | 0 | 0 | 0 | 0 |

Below is a list of problems that people sometimes have in response to a very stressful experience. Please read each problem carefully and then indicate how much you have been bothered by that problem in the past month.

In the **past month**, how much were you bothered by:

| | Not at all | A little bit | Moderately | Quite a bit | Extremely |
|---|---|---|---|---|---|
| Having strong negative feelings such as fear, horror, anger, guilt, or shame? | 0 | 0 | 0 | 0 | 0 |
| Loss of interest in activities that you used to enjoy? | 0 | $\circ$ | $\circ$ | 0 | $\circ$ |
| Feeling distant or cut off from other people? | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Trouble experiencing positive feelings (for example, being unable to feel happiness or have loving feelings for people close to you)? | 0 | $\circ$ | 0 | 0 | 0 |
| Irritable behavior, angry outbursts, or acting aggressively? | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| Taking too many risks or doing things that could cause you harm? | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| Being "superalert" or watchful or on guard? | 0 | | $\circ$ | 0 | $\circ$ |
| Feeling jumpy or easily startled? | 0 | $\circ$ | $\circ$ | 0 | $\circ$ |
| Having difficulty concentrating? | 0 | | $\circ$ | $\circ$ | $\circ$ |
| Trouble falling or staying asleep? | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |

#### BMI (Body Mass Index)

| What is your height (in feet and inches)? |
|---|
| What is your weight (in pounds)? (If pregnant, please use pre-pregnancy weight.) |
| RQoL (Health Related Quality of Life) |
| Would you say that in general your health is — |
| Excellent |
| ○ Very good |
| Good |
| ○ Fair |
| O Poor |
| On't know/not sure |
| Now thinking about your <b>physical health</b> , which includes physical illness and injury, for how many days during the <b>past 30 days</b> was your physical health <b>not good</b> ? |
| Now thinking about your <u>mental health</u> , which includes stress, depression, and problems with |
| emotions, for how many days during the past 30 days was your mental health not good? |

| During the <u>past 30 days</u> , for about how many days did <u>poor physical or mental health</u> keep you from doing your usual activities, such as self care, work, or recreation? |
|---|

## AD (Autoimmune Disease)

| ○ No ○ Yes, I have been diagnosed with: | <u>sease</u> ?<br>.g., rheumatoid ar | or other health profe<br>hritis, hashimoto's dis<br>upus erythematosus) |
|---|---|---|
| Yes, I have been diagnosed with: | No | |
| | Yes, I have been diagnosed | with: |

## PHQ-15 (Somatic Symptoms Survey)

| How much have you been bothered by any of the following problems? | | | |
|---|---|---|---|
| | Not bothered at all | Bothered a little | Bothered a lot |
| Stomach pain | 0 | 0 | 0 |
| ack pain | 0 | 0 | 0 |
| ain in your arms, legs, or joints (knees, hips, etc.) | 0 | $\circ$ | 0 |
| lenstrual cramps or other problems with your periods [Women only] | 0 | 0 | 0 |
| leadaches | 0 | 0 | 0 |
| hest pain | 0 | 0 | 0 |
| Dizziness | 0 | 0 | 0 |
| ainting spells | 0 | 0 | 0 |
| eeling your heart pound or race | 0 | 0 | 0 |
| hortness of breath | 0 | 0 | 0 |
| ain or problems during sexual intercourse | 0 | 0 | 0 |
| constipation, loose bowels, or diarrhea | 0 | 0 | 0 |
| lausea, gas, or indigestion | 0 | $\circ$ | 0 |
| Feeling tired or having low energy | 0 | 0 | 0 |

| | $\circ$ | | 0 | | 0 |
|---|---|---|---|---|---|
| T (Alcohol) | | | | | |
| he following are questions about your alcohol use i | n the <u>pa</u> | ıst 12 mo | nths. | | |
| How often do you have one drink containing alcoho | 1? | | | | |
| Never | | | | | |
| Monthly or less | | | | | |
| 2-4 times a month | | | | | |
| 2-3 times a week | | | | | |
| 4 or more times a week | | | | | |
| 1 or 2<br>3 or 4 | a typica | l day whe | n you are | e drinkinç | g? |
| 1 or 2 | a typica | l day whe | n you are | e drinking | <b>]</b> ? |
| 3 or 4<br>5 or 6<br>7 to 9 | a typica | I day whe | n you are | e drinking | |
| 1 or 2<br>3 or 4<br>5 or 6<br>7 to 9 | a typica | I day whe | n you are | e drinking<br>Weekly | Daily or<br>almost<br>daily |
| 1 or 2 3 or 4 5 or 6 7 to 9 10 or more ow often do you have four or more drinks on one occasion? | | Less than | | | Daily or almost |
| 1 or 2 3 or 4 5 or 6 7 to 9 10 or more ow often do you have four or more drinks on one occasion? ow often during the last year have you found that you are not able to stop | | Less than | | | Daily or almost |
| 1 or 2 3 or 4 5 or 6 7 to 9 10 or more ow often do you have four or more drinks on one occasion? ow often during the last year have you found that you are not able to stop inking once you have started? ow often during the last year have you failed to do what was normally | | Less than | | | Daily or almost |
| 1 or 2 3 or 4 5 or 6 7 to 9 10 or more ow often do you have four or more drinks on one occasion? ow often during the last year have you found that you are not able to stop inking once you have started? ow often during the last year have you failed to do what was normally pected from you because of drinking? ow often during the last year have you needed a first drink in the morning to | | Less than | | | Daily or almost |
| 1 or 2<br>3 or 4<br>5 or 6<br>7 to 9 | | Less than | | | Daily or almost |

| In the past 12 months | | | |
|---|---|---|---|
| | No | Yes, but not in the last year | Yes, during the last year |
| Have you or someone else been injured as a result of your drinking? | 0 | 0 | 0 |
| Has a relative or friend or doctor or health worker been concerned about your drinking or suggested you cut down? | 0 | 0 | 0 |

## TAPS (Substance Use)

| The following are questions about other substance use. | | | | | |
|---|---|---|---|---|---|
| In the past 12 months, how often have you | | | | | |
| | Never | Less than monthly | Monthly | Weekly | Daily or<br>almost<br>daily |

# Used any prescription medications just for the feeling, more than prescribed or that were not prescribed for you? Used any other drugs including cocaine or crack, heroin, meth, hallucinogens, ecstasy/MDMA?

## JSS (Sleep Disturbance)

Used marijuana?

| In the <b>past month</b> , did you | | | | | | |
|---|---|---|---|---|---|---|
| | Not at all | 1-3 days | 4-7 days | 8-14 days | 15-21 days | 22-31 days |
| Have trouble falling asleep? | 0 | 0 | 0 | 0 | 0 | 0 |
| Wake up several times per night? | 0 | 0 | 0 | 0 | 0 | $\circ$ |
| Have trouble staying asleep (including waking far too early)? | 0 | 0 | 0 | 0 | 0 | 0 |
| Wake up after your usual amount of sleep feeling tired and worn out? | 0 | 0 | 0 | 0 | 0 | 0 |
| | I | | | | | |

## GAD-7 (Anxiety)

Over the last two weeks, how often have you been bothered by the following problems? Indicate how often you have experienced... More than half the Not at all Several days days Nearly every day Feeling nervous, anxious or on edge. 0 0 0 0 Not being able to stop or control worrying. Worrying too much about different things. Trouble relaxing. Being so restless that it is hard to sit still. Becoming easily annoyed or irritable. Feeling afraid as if something awful might happen.

#### PHQ-8 (Depression)

Over the <u>last two weeks</u>, how often have you been bothered by any of the following problems?

Indicate how often any of the following problems have bothered you.

| | Not at all | Several days | More than half the days | Nearly every day |
|---|---|---|---|---|
| Little interest or pleasure doing things. | 0 | 0 | 0 | 0 |
| Feeling down, depressed, or hopeless. | 0 | 0 | 0 | 0 |
| Trouble falling or staying asleep, or sleeping too much. | 0 | $\circ$ | 0 | 0 |
| Feeling tired or having little energy. | 0 | 0 | 0 | |
| Poor appetite or overeating. | 0 | $\circ$ | $\circ$ | |
| Feeling bad about yourself - or that you are a failure or have let yourself or your family down. | 0 | 0 | $\circ$ | $\circ$ |
| Trouble concentrating on things, such as reading the newspaper or watching television. | 0 | 0 | $\circ$ | 0 |
| Moving or speaking so slowly that other people could have noticed. Or the opposite - being so fidgety or restless that you have been moving around a lot more than usual. | 0 | 0 | 0 | 0 |

#### MHS (Mental Health Specialist)

In the past month, have you talked to a mental health specialist, such as a psychiatrist, psychologist, or specially trained social worker, about emotional problems, your nerves, or the
| way you were feeling or behaving? |
|-----------------------------------|
| ○ No |
| ○ Yes |

# IRI (Empathy)

| | l _ | | | | _ |
|---|---|---|---|---|---|
| | Does not describe me well | 2 | 3 | 4 | Does<br>describe<br>me well |
| I daydream and fantasize, with some regularity, about things that might happen to me. | 0 | 0 | 0 | 0 | 0 |
| I often have tender, concerned feelings for people less fortunate than me. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I sometimes find it difficult to see things from the "other person's" point of view. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Sometimes I don't feel very sorry for other people when they are having problems. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I really get involved with the feelings of the characters in a novel. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| In emergency situations, I feel apprehensive and ill-at-ease. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I am usually objective when I watch a movie or play, and I don't often get completely caught up in it. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I try to look at everybody's side of a disagreement before I make a decision. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| When I see someone being taken advantage of, I feel kind of protective towards them. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I sometimes feel helpless when I am in the middle of a very emotional situation. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I sometimes try to understand my friends better by imagining how things look from their perspective. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Becoming extremely involved in a good book or movie is somewhat rare for me. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| When I see someone get hurt, I tend to remain calm. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Other people's misfortunes do not usually disturb me a great deal. | 0 | 0 | 0 | 0 | 0 |

| Does not describe me well | 2 | 3 | 4 | Does<br>describe<br>me well |
|---|---|---|---|---|
| 0 | 0 | 0 | 0 | 0 |
| 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| 0 | 0 | $\circ$ | 0 | $\circ$ |
| | describe | describe | describe | describe |

| Lwould describe myself as a protty self bearted person | | $\bigcirc$ | 0 | | |
|---|---|---|---|---|---|
| I would describe myself as a pretty soft-hearted person. | 0 | 0 | 0 | 0 | 0 |
| When I watch a good movie, I can very easily put myself in the place of a leading character. | 0 | 0 | 0 | 0 | 0 |
| I tend to lose control during emergencies. | 0 | 0 | 0 | 0 | 0 |
| When I'm upset at someone, I usually try to "put myself in his shoes" for a while. | 0 | 0 | 0 | 0 | 0 |
| When I am reading an interesting story or novel, I imagine how I would feel if the events in the story were happening to me. | 0 | 0 | 0 | 0 | 0 |
| When I see someone who badly needs help in an emergency, I go to pieces. | 0 | 0 | 0 | 0 | 0 |
| Before criticizing somebody, I try to imagine how I would feel if I were in their place. | 0 | 0 | 0 | 0 | 0 |
| BRFSS Adverse Childhood Experiences (ACEs) | | | | | |
| Next are some questions about events that happened <u>during your</u> information will allow us to better understand problems that may occ help others in the future. <u>Trigger warning</u> . This is a sensitive topic uncomfortable with these questions. Please keep in mind that you can do not want to answer. All questions refer to the time period before Now, looking back before you were 18 years of age | ur early<br>and som<br>an skip a | in<br>ne p<br>any | life a<br>eopl<br>que: | and m<br>le may<br>stion | / feel<br>you |
| | | | | | Don't<br>know/not |
| | | | No | o Yes | sure |
| Did you live with anyone who was depressed, mentally ill, or suicidal? | | | | | 0 |
| Did you live with anyone who were a problem drinker or electric? | | | | | |
| Did you live with anyone who was a problem drinker or alcoholic? | | | | | |
| Did you live with anyone who used illegal street drugs or who abused prescription medications? | : | 0 | 0 | 0 | 0 |
| | ional facility | ? | 0 | 0 0 | 0 |
| Did you live with anyone who used illegal street drugs or who abused prescription medications? | ional facility | ? | | 0 0 | 0 |
| Did you live with anyone who used illegal street drugs or who abused prescription medications? Did you live with anyone who served time or was sentenced to serve time in a prison, jail, or other correct | | | Yes | Don't know/not sure | Parents not married |
| Did you live with anyone who used illegal street drugs or who abused prescription medications? Did you live with anyone who served time or was sentenced to serve time in a prison, jail, or other correct | | | | know/not | not |
| Did you live with anyone who used illegal street drugs or who abused prescription medications? Did you live with anyone who served time or was sentenced to serve time in a prison, jail, or other correct Now, looking back before you were 18 years of age | | | | know/not | not |
| Did you live with anyone who used illegal street drugs or who abused prescription medications? Did you live with anyone who served time or was sentenced to serve time in a prison, jail, or other correct Now, looking back before you were 18 years of age | | | | know/not | not |

Qualtrics Survey Software 8/6/19, 7:38 PM How often did your parents or adults in your home ever slap, hit, kick, punch or beat each other up? How often did a parent or adult in your home ever hit, beat, kick, or physically hurt you in any way? Do not include spanking. How often did a parent or adult in your home ever swear at you, insult you, or put you down? How often did anyone at least 5 years older than you or an adult, ever touch you sexually? How often did anyone at least 5 years older than you or an adult, try to make you touch sexually? How often did anyone at least 5 years older than you or an adult, force you to have sex? BRS (Resilience)

| | Strongly disagree | Disagree | Neutral | Agree | Strongly<br>agree |
|---|---|---|---|---|---|
| tend to bounce back quickly after hard times. | 0 | 0 | 0 | 0 | 0 |
| have a hard time making it through stressful events. | 0 | 0 | 0 | 0 | 0 |
| t does not take me long to recover from a stressful event. | 0 | 0 | 0 | 0 | 0 |
| is hard for me to snap back when something bad happens. | 0 | 0 | 0 | 0 | 0 |
| usually come through difficult times with little trouble. | 0 | 0 | 0 | 0 | 0 |
| tend to take a long time to get over set-backs in my life. | 0 | 0 | 0 | 0 | 0 |

## ECR-RS (Experiences in Close Relationships - Relationship Structures)

Please read each of the following statements and rate the extent to which you believe each statement best describes your feelings about close relationships in general.

| | Strongly disagree | 2 | 3 | 4 | 5 | 6 | Strongly agree |
|---|---|---|---|---|---|---|---|
| It helps to turn to people in times of need. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| I usually discuss my problems and concerns with others. | 0 | 0 | $\circ$ | $\circ$ | $\circ$ | 0 | $\circ$ |
| I talk things over with people. | 0 | $\circ$ | $\circ$ | 0 | 0 | $\circ$ | |
| I find it easy to depend on others. | 0 | $\circ$ | $\circ$ | 0 | 0 | $\circ$ | 0 |
| I don't feel comfortable opening up to others. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| I prefer not to show others how I feel deep down. | 0 | $\circ$ | 0 | 0 | 0 | $\circ$ | 0 |
| I often worry that other people do not really care for me. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| I'm afraid that other people may abandon me. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

| I worry that others won't care about me as much as I care about them. |
|-----------------------------------------------------------------------|
|-----------------------------------------------------------------------|

# MAIA (Interoceptive Awareness)

Qualtrics Survey Software

| Please indicate how often each statement applies to you generally in daily life: | | | | | | |
|---|---|---|---|---|---|---|
| | Never | 1 | 2 | 3 | 4 | Always |
| When I am tense I notice where the tension is ocated in my body. | 0 | 0 | 0 | 0 | 0 | 0 |
| notice when I am uncomfortable in my body. | 0 | $\circ$ | 0 | 0 | $\circ$ | 0 |
| notice where in my body I am comfortable. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | 0 |
| notice changes in my breathing, such as whether it lows down or speeds up. | 0 | 0 | 0 | 0 | 0 | 0 |
| gnore physical tension or discomfort until they ecome more severe. | 0 | 0 | 0 | 0 | $\circ$ | $\circ$ |
| distract myself from sensations of discomfort. | 0 | 0 | 0 | 0 | 0 | 0 |
| /hen I feel pain or discomfort, I try to power rough it. | 0 | $\circ$ | 0 | 0 | $\circ$ | 0 |
| try to ignore pain. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | 0 |
| oush feelings of discomfort away by focusing on omething. | 0 | 0 | 0 | 0 | 0 | $\circ$ |
| When I feel unpleasant body sensations, I occupy<br>hyself with something else so I don't have to feel<br>hem. | 0 | 0 | 0 | 0 | 0 | 0 |
| /hen I feel physical pain, I become upset. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | 0 |
| start to worry that something is wrong if I feel any scomfort. | 0 | 0 | 0 | 0 | $\circ$ | $\circ$ |

| Below you will find a list of statemen | nts. | | | | | |
|---|---|---|---|---|---|---|
| Please indicate how often each state | ement appl | ies to you | generally | in daily l | ife: | |
| | Never | 1 | 2 | 3 | 4 | Always |
| I can notice an unpleasant body sensation without worrying about it. | 0 | 0 | 0 | 0 | 0 | 0 |
| I can stay calm and not worry when I have feelings of discomfort or pain. | 0 | 0 | $\circ$ | $\circ$ | 0 | 0 |
| When I am in discomfort or pain I can't get it out of my mind. | 0 | 0 | 0 | 0 | 0 | $\circ$ |
| I can pay attention to my breath without being distracted by things happening around me. | 0 | 0 | 0 | $\circ$ | 0 | 0 |
| I can maintain awareness of my inner bodily sensations even when there is a lot going on around | | | | | | |

| me. | 0 | 0 | 0 | 0 | 0 | $\circ$ |
|---|---|---|---|---|---|---|
| When I am in conversation with someone, I can pay attention to my posture. | 0 | 0 | 0 | 0 | 0 | $\circ$ |
| I can return awareness to my body if I am distracted. | 0 | $\circ$ | $\circ$ | 0 | $\circ$ | $\circ$ |
| I can refocus my attention from thinking to sensing my body. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 | 0 |
| I can maintain awareness of my whole body even when a part of me is in pain or discomfort. | 0 | $\circ$ | 0 | 0 | 0 | $\circ$ |
| I am able to consciously focus on my body as a whole. | 0 | $\circ$ | 0 | 0 | 0 | $\circ$ |
| I notice how my body changes when I am angry. | 0 | $\circ$ | $\circ$ | 0 | $\circ$ | 0 |
| When something is wrong in my life I can feel it in my body. | 0 | $\circ$ | 0 | 0 | 0 | $\circ$ |
| I notice that my body feels different after a peaceful experience. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 | $\circ$ |

| Below you will find a list of statements. | | | | | | |
|---|---|---|---|---|---|---|
| Please indicate how often each stat | ement appl | ies to you | generally | in daily l | ife: | |
| | Never | 1 | 2 | 3 | 4 | Always |
| notice that my breathing becomes free and easy when I feel comfortable. | 0 | 0 | 0 | 0 | 0 | 0 |
| notice how my body changes when I feel happy / oyful. | 0 | 0 | 0 | 0 | 0 | $\circ$ |
| When I feel overwhelmed I can find a calm place inside. | 0 | 0 | 0 | 0 | 0 | $\circ$ |
| When I bring awareness to my body I feel a sense of calm. | 0 | 0 | 0 | 0 | 0 | 0 |
| can use my breath to reduce tension. | 0 | | $\circ$ | $\circ$ | | $\circ$ |
| When I am caught up in thoughts, I can calm my mind by focusing on my body/breathing. | 0 | 0 | 0 | 0 | $\circ$ | 0 |
| listen for information from my body about my emotional state. | 0 | $\circ$ | 0 | 0 | 0 | 0 |
| When I am upset, I take time to explore how my body feels. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 | $\circ$ |
| listen to my body to inform me about what to do. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| am at home in my body. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | 0 |
| feel my body is a safe place. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I trust my body sensations. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |

# FFMQ (Five Facets of Mindfulness)

Qualtrics Survey Software

Choose the best response that describes your opinion of what is generally true for you.

| | Never<br>or very<br>rarely<br>true | Rarely<br>true | Sometimes true | Often<br>true | Very<br>often or<br>always<br>true |
|---|---|---|---|---|---|
| When I'm walking, I deliberately notice the sensations of my body moving. | 0 | 0 | 0 | 0 | 0 |
| I'm good at finding words to describe my feelings. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I criticize myself for having irrational or inappropriate emotions. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| I perceive my feelings and emotions without having to react to them. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| When I do things, my mind wanders off and I'm easily distracted. | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| When I take a shower or bath, I stay alert to the sensations of water on my body. | $\circ$ | $\circ$ | 0 | $\circ$ | $\circ$ |
| I can easily put my beliefs, opinions, and expectations into words. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I don't pay attention to what I'm doing because I'm daydreaming, worrying, or otherwise distracted. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| I watch my feelings without getting lost in them. | $\circ$ | $\circ$ | 0 | $\circ$ | $\circ$ |
| I tell myself I shouldn't be feeling the way I'm feeling. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| I notice how foods and drinks affect my thoughts, bodily sensations, and emotions. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| It's hard for me to find the words to describe what I'm thinking. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I am easily distracted. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Please select 'Very often' for this response. | 0 | 0 | 0 | 0 | 0 |

| Choose the best response that describes your opinion of what | is gene | erally | true for y | ou. | |
|---|---|---|---|---|---|
| | Never<br>or very<br>rarely<br>true | Rarely<br>true | Sometimes true | Often<br>true | Very<br>often or<br>always<br>true |
| I believe some of my thoughts are abnormal or bad and I shouldn't think that way. | 0 | 0 | 0 | 0 | 0 |
| I pay attention to sensations, such as the wind in my hair or sun on my face. | 0 | $\circ$ | | $\circ$ | $\circ$ |
| I have trouble thinking of the right words to express how I feel about things. | 0 | $\circ$ | | $\circ$ | $\circ$ |
| I make judgments about whether my thoughts are good or bad. | 0 | $\circ$ | | $\circ$ | $\circ$ |
| I find it difficult to stay focused on what's happening in the present. | 0 | $\circ$ | | $\circ$ | $\circ$ |
| When I have distressing thoughts or images, I "step back" and am aware of the thought or image without getting taken over by it. | 0 | 0 | $\circ$ | $\circ$ | 0 |
| I pay attention to sounds, such as clocks ticking, birds chirping, or cars passing. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| In difficult situations, I can pause without immediately reacting. | 0 | $\circ$ | | $\circ$ | $\circ$ |
| When I have a sensation in my body, it's difficult for me to describe it because I can't find the right words. | 0 | 0 | $\circ$ | $\circ$ | $\circ$ |
| It seems I am "running on automatic" without much awareness of what I'm doing. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| When I have distressing thoughts or images, I feel calm soon after. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| I tell myself that I shouldn't be thinking the way I'm thinking. | 0 | $\circ$ | | $\circ$ | $\circ$ |
| I notice the smells and aromas of things. | 0 | 0 | $\circ$ | 0 | $\circ$ |

| | Never<br>or very<br>rarely<br>true | Rarely<br>true | Sometimes true | Often<br>true | Very<br>often<br>alway<br>true |
|---|---|---|---|---|---|
| ven when I'm feeling terribly upset, I can find a way to put it into words. | 0 | 0 | 0 | 0 | 0 |
| ush through activities without being really attentive to them. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| hen I have distressing thoughts or images I am able just to notice them without reacting. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| hink some of my emotions are bad or inappropriate and I shouldn't feel them. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| notice visual elements in art or nature, such as colors, shapes, textures, or patterns of light and shadow. | 0 | 0 | $\circ$ | 0 | 0 |
| y natural tendency is to put my experiences into words. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| hen I have distressing thoughts or images, I just notice them and let them go. | 0 | $\circ$ | 0 | $\circ$ | 0 |
| to jobs or tasks automatically without being aware of what I'm doing. | 0 | $\circ$ | 0 | $\circ$ | 0 |
| hen I have distressing thoughts or images, I judge myself as good or bad, depending what e thought/image is about. | 0 | 0 | $\circ$ | 0 | 0 |
| pay attention to how my emotions affect my thoughts and behavior. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| can usually describe how I feel at the moment in considerable detail. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| ind myself doing things without paying attention. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| disapprove of myself when I have irrational ideas. | 0 | 0 | 0 | 0 | 0 |
| Trauma Exposure and Training Questions) Overall, how much of your work involves (directly or indirectly) | engag | ina wi | th trauma | ıtized | |

How much training have you received on primary or secondary trauma (including topics like vicarious trauma, secondary traumatic stress, burnout, and moral distress)?

A great deal

A moderate amount

A littleNone at all

O A lot

| | A moderate amount |
|---|---|
| | A little |
| | None at all |
| | Altogether, how effective were your trainings on primary or secondary trauma (including topics like vicarious trauma, secondary traumatic stress, burnout, and moral distress)? |
| | Extremely effective |
| | O Very effective |
| | Moderately effective |
| | ◯ Slightly effective |
| | Not effective at all |
| | Do you want more training on secondary trauma (including topics like vicarious trauma, secondary traumatic stress, burnout, and moral distress)? |
| | Oefinitely yes |
| | Probably yes |
| | Might or might not |
| | O Probably not |
| | Definitely not |
| E | (Feedback) |
| | Are there any factors affecting your answers that we should know about (e.g., a health issue or language barrier)? |
| | Please provide any other feedback you would like to share. |

| Identifiers |
|---|
| Thank you for participating in our survey. We would like to email you an Amazon.com eGift Card. To do so, we need you to complete the following questions. Please allow one week for us to email you the eGift Card. Thanks for your patience with us! |
| What is your first name? |
| What is your last name? |
| What is your phone number (e.g., XXX-XXX-XXXX)? |
| What is your email address? (This is where we will send your e-gift card.) |

| Please verify your email address. |
|-----------------------------------|

#### Consent, MSU Students

#### Hello!

This survey has been developed by Associate Professors from Montana State University to study secondary trauma.

The purpose of this study is to better understand the personal histories and experiences of victim service providers, or those considering becoming victim service providers, in Montana.

Any insights you could offer are greatly appreciated!

Before we begin, however, we need to review this consent form. This insures that your rights are protected as a participant this study.

Kelly Knight, PhD Principal Investigator

#### Questions? We have answers:

#### Why am I being asked to participate?

You are being asked to participate in a research study because of your current or future involvement in, or knowledge of, services in your area.

#### Why is this research being done?

This survey is being conducted to evaluate a new educational program. The program is intended to teach people strategies for managing the negative consequences of secondary trauma. Your participation will help us better understand how the personal histories and experiences of service providers impact their work and mental and physical health.

#### How long will it take me to participate?

This survey should take approximately 30-45 minutes to complete.

#### Will I be compensated for participation?

No, you will not be compensated for your involvement. You will, however, receive an e-gift card if you complete this survey a third time.

#### What will I be asked to do?

Your participation in this research is voluntary and completely your choice. It will in no way impact your grade in this class or your relationship with your professors. If you agree, you

will be asked to answer a number of questions about your personal history, your work, your physical and psychological health, and your resilience. You will also be asked to complete some basic demographic questions. You can choose to not answer questions you do not want to answer. Also, you can stop at any time with no consequences.

#### Are there any benefits to me if I participate in this study?

This study is of no direct benefit to you. However, the information gained will inform the development of a data-driven intervention to lessen the impacts of secondary trauma on service providers.

### Will my information be kept private?

Everything you tell us will be kept confidential. Your answers will be separated from your name and contact information (which will be used for tracking purposes only).

All data collected will be secured on a password-protected and firewalled computer in a locked office on Montana State University's campus or stored on a secure server. No one but the official research staff will have access to the information. Your results will be grouped with other participants' data when results of this study is published. Your identity will remain anonymous.

An exception to confidentiality is the indication of imminent harm to yourself or others.

## Who should I contact if I have questions?

You can contact the principal investigator about the study: Kelly E. Knight, PhD, (406) 994-7224, kelly.knight3@montana.edu. They can also be reached by mail at: Montana State University, Department of Sociology and Anthropology, PO Box 172380, Bozeman, MT, 59817.

In addition, you can contact MSU's institutional review board chairperson: Mark Quinn, PhD, (406) 994-4747, mquinn@montana.edu. He can also be reached by mail at Montana State University, IRB, PO BOX 173610, Bozeman, MT, 59817.

#### What happens if I change my mind?

Participation is strictly voluntary and you can stop at any time. Participation or non-participation will not affect your current or future relationship with Montana State University.

#### Are there any risks to me if I participate in this study?

We do not foresee any significant physical or psychological risks as a result of your participation. However, some of the questions are personal and may provoke an emotional response. Below is a list of resources should you be worried or need support after the survey.

#### Resource List:

1. Montana Suicide Prevention Lifeline: (800) 273-8255

- 2. MSU Voice Center: (406) 994-7069
- 3. Counseling and Psychological Services, MSU: (406) 994-4531
- 4. HELP Center Crisis and Referral Line: (406) 586-3333 or just dial 2-1-1
- 5. Haven Domestic Violence Program: (406) 586-4111
- 6. Alcohol and Drug Services of Gallatin County: (406) 586-5493
- 7. Bozeman Health Deaconess Hospital: (406) 414-5000
- 8. Bridger Care, Reproductive & Sexual Healthcare & Education: (406) 587-0681
- 9. Child and Family Services: (866) 820-5437
- 10. Gallatin Valley Mental Health Center: (406) 556-6500

#### **ELECTRONIC CONSENT:**

- You voluntarily agree to participate.
- You are 18 years of age or older.
- Agree

## BDS (Basic Demographics, Student)

| What is yo | our sex/gender? |
|------------|-----------------|
| Female | |
| O Male | |
| Other | |

| What is your current marital status? |
|---------------------------------------|
| ○ Married |
| Living with partner (but not married) |
| O Divorced/separated |

| Single | |
|---|---|
| Widowed | |
| Other | |
| Culci | |
| What race do you consid | er yourself? Check all that apply. |
| American Indian | |
| Alaskan Native | |
| Asian | |
| Black or African American | |
| Hispanic or Latino | |
| <ul> <li>Native Hawaiian, Other Pacific Is</li> </ul> | ander |
| Other | |
| What is your ago? | |
| What is your age? | |
| What is your age? | |
| What is your age? | |
| What is your age? | |
| • | |
| What is your major? | |
| What is your age? What is your major? Major: Second major (if applicable): | |
| What is your major? Major: | |
| What is your major? Major: Second major (if applicable): | 5? |
| What is your major? Major: Second major (if applicable): | 5? |
| What is your major? Major: Second major (if applicable): What is your class statu | s? |
| What is your major? Major: Second major (if applicable): What is your class statu | 5? |

| Graduate student |
|---------------------------------------------------------|
| Professional student |
| Continuing education student |
| How many hours/week do you work for pay OFF campus? |
| How many hours/week do you work for pay ON campus? |
| How many hours/week of volunteer work? |
| Do you consider yourself to be a veteran? Yes No |
| Do you consider yourself to be an NCAA athlete? Yes No |

| No | | | | | | | |
|---|---|---|---|---|---|---|---|
| O ADHD/ADD | | | | | | | |
| <ul><li>Learning disability</li></ul> | | | | | | | |
| Physical disability | | | | | | | |
| Psychological disability | | | | | | | |
| Traumatic brain injury | | | | | | | |
| Other: | | | | | | | |
| BI-S (Maslach Burnout Inventory - St | | - | Diagon | | | | |
| Below are 17 statements of universit decide if you ever feel this way about indicate how often you feel it by indifeel that way. | it your ac | cademic | work. If | you have | had this | s feeling | ], |
| | Never | A few<br>times a<br>year or<br>less | Once a<br>month or<br>less | A few times<br>a month | Once a<br>week | A few times a week | Every day |
| I feel emotionally drained by my studies. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| I feel used up at the end of the day at the university. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I feel tired when I get up in the morning and have to face another day at the university. | 0 | $\circ$ | 0 | 0 | $\circ$ | 0 | 0 |
| Attending classes all day is really a strain for me. | 0 | 0 | 0 | 0 | $\circ$ | 0 | 0 |
| I can effectively solve the problems that arise in my studies. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| I feel burned out from my studies. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| I feel I am making an effective contribution in class. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| I have become less interested in my studies since my enrollment. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Copyright ©1996 Wilmar B. Schaufeli, Michael<br>media. Published by Mind Garden, Inc., www.m | P. Leiter, C<br>nindgarden. | com | aslach & Si | usan E. Jack | son. All ri | ghts reser | ved in all |
| On this page are statements of job-r decide if you ever feel this way abou | | | lease re | ad each s | tatemer | nt carefu | Ily and |
| A | A few times a | Once a | A few tim | ies a | A fe | w times a | |

8/6/19, 7:37 PM Qualtrics Survey Software Never year or less month or less month Once a week week Everyday I have become less enthusiastic about my studies. In my opinion, I am a good student. I feel exhilarated when I accomplish something at the university. I have accomplished many worthwhile things in my studies. I just want to get my work done and not be bothered. I have become more cynical about whether my university work contributes to anything. I doubt the significance of my studies While working at the university, I feel confident that I am effective at getting things done. Copyright @1996 Wilmar B. Schaufeli, Michael P. Leiter, Christina Maslach & Susan E. Jackson. All rights reserved in all media. Published by Mind Garden, Inc., www.mindgarden.com MBI-GS (Maslach Burnout Inventory - General Student Version) Do you currently work (for a wage or as a volunteer)? Yes, I currently work either for a wage or as a volunteer. No, I do not currently work or volunteer. On this page are statements of job-related feelings. Please read each statement carefully and decide if you ever feel this way about your job. A few times a Once a A few year or month or A few times Once a times a Every day Never a month week week less less I feel emotionally drained from my work.  $\bigcirc$ I feel used up at the end of the workday.

I feel tired when I get up in the morning and have to

face another day on the job.

| Working all day is really a strain for me. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
|---|---|---|---|---|---|---|---|
| I can effectively solve the problems that arise in my work. | 0 | 0 | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I feel burned out from my work. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| I feel I am making an effective contribution to what this organization does. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I have become less interested in my work since I started this job. | 0 | 0 | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| | I | | | | | | |
| Copyright ©1996 Wilmar B. Schaufeli, Michael | | | | | | | |

On this page are statements of job-related feelings. Please read each statement carefully and decide if you ever feel this way about your job.

| | Never | A few times a<br>year or less | Once a month or less | A few times a month | Once a week | A few times a week | Every day |
|---|---|---|---|---|---|---|---|
| I have become less enthusiastic about my work. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| In my opinion, I am good at my job. | $\circ$ | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I feel exhilarated when I accomplish something at work. | $\circ$ | 0 | 0 | 0 | 0 | $\circ$ | $\circ$ |
| I have accomplished many worthwhile things in this job. | $\circ$ | 0 | $\circ$ | 0 | $\circ$ | $\circ$ | $\circ$ |
| I just want to do my job and not be bothered. | $\circ$ | 0 | $\circ$ | 0 | $\circ$ | $\circ$ | $\circ$ |
| I have become more cynical about whether my work contributes anything. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| I doubt the significance of my work. | $\circ$ | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| At my work, I feel confident that I am effective at getting things done. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

Copyright ©1996 Wilmar B. Schaufeli, Michael P. Leiter, Christina Maslach & Susan E. Jackson. All rights reserved in all media. Published by Mind Garden, Inc., www.mindgarden.com

## STSS (Secondary Traumatic Stress Scale)

Qualtrics Survey Software

The following is a list of statements made by persons who have been impacted by their work with traumatized clients (or other potentially traumatized populations, e.g., patients, students, customers, or anyone to whom you provide services).

In the **past seven** days, how frequently was the statement true for you:

| | Never | Rarely | Occasionally | Often | Very often |
|---|---|---|---|---|---|
| I felt emotionally numb. | 0 | 0 | 0 | 0 | 0 |
| My heart started pounding when I thought about my work with clients. | 0 | 0 | 0 | $\circ$ | 0 |
| It seemed as if I was reliving the trauma(s) experienced by my client(s). | 0 | 0 | 0 | $\circ$ | $\circ$ |
| I had trouble sleeping. | 0 | $\circ$ | 0 | $\circ$ | |
| I felt discouraged about the future. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Reminders of my work with clients upset me. | 0 | $\circ$ | 0 | $\circ$ | |
| I had little interest in being around others. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| I felt jumpy. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I was less active than usual. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I thought about my work with clients when I didn't intend to. | 0 | $\circ$ | 0 | $\circ$ | |
| I had trouble concentrating. | 0 | $\circ$ | 0 | $\circ$ | |
| I avoided people, places, or things that reminded me of my work with clients. | 0 | $\circ$ | 0 | $\circ$ | |
| I had disturbing dreams about my work with clients. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I wanted to avoid working with some clients. | 0 | $\circ$ | 0 | $\circ$ | |
| I was easily annoyed. | 0 | $\circ$ | 0 | $\circ$ | |
| I expected something bad to happen. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I noticed gaps in my memory about client sessions. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Please select 'Very often' for this response. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| | • | | | | |

## PCL-5 (PTSD)

Below is a list of problems that people sometimes have in response to a very stressful experience. Please read each problem carefully and then indicate how much you have been bothered by that problem in the past month.

In the **past month**, how much were you bothered by:

| | Not at all | A little bit | Moderately | Quite a bit | Extremely |
|---|---|---|---|---|---|
| Repeated, disturbing, and unwanted memories of the stressful experience? | 0 | 0 | 0 | 0 | 0 |
| Repeated, disturbing dreams of the stressful experience? | 0 | 0 | 0 | $\circ$ | 0 |
| Suddenly feeling or acting as if the stressful experience were actually happening again (as if you were actually back there reliving it)? | 0 | 0 | $\circ$ | 0 | $\circ$ |
| Feeling very upset when something reminded you of the stressful experience? | 0 | 0 | 0 | 0 | 0 |

| | | | | | 8/6/19, |
|---|---|---|---|---|---|
| Having strong physical reactions when something reminded you of the stressful experience (for example, heart pounding, trouble breathing, sweating)? | 0 | 0 | 0 | 0 | 0 |
| Avoiding memories, thoughts, or feelings related to the stressful experience? | 0 | 0 | 0 | 0 | 0 |
| Avoiding external reminders of the stressful experience (for example, people, places, conversations, activities, objects, or situations)? | 0 | 0 | 0 | 0 | 0 |
| Trouble remembering important parts of the stressful experience? | 0 | 0 | 0 | 0 | 0 |
| Having strong negative beliefs about yourself, other people, or the world (for example, having thoughts such as: I am bad, there is something seriously wrong with me, no one can be trusted, the world is completely dangerous)? | 0 | 0 | 0 | 0 | 0 |
| Blaming yourself or someone else for the stressful experience or what happened after it? | 0 | 0 | 0 | 0 | 0 |
| experience. Please read each problem carefully bothered by that problem in the past month. In the <b>past month</b> , how much were you bothered. | ed by: | | | | |
| Having strong negative feelings such as fear, horror, anger, guilt, or | Not at all | A little bit | Moderately | Quite a bit | Extremely |
| shame? | 0 | 0 | 0 | 0 | 0 |
| Loss of interest in activities that you used to enjoy? | 0 | 0 | 0 | $\circ$ | 0 |
| | 0 | $\circ$ | 0 | 0 | 0 |
| Feeling distant or cut off from other people? | | | | | |
| Trouble experiencing positive feelings (for example, being unable to feel | 0 | $\circ$ | 0 | 0 | 0 |
| Trouble experiencing positive feelings (for example, being unable to feel happiness or have loving feelings for people close to you)? | 0 | 0 | 0 | 0 | 0 |
| Trouble experiencing positive feelings (for example, being unable to feel happiness or have loving feelings for people close to you)? Irritable behavior, angry outbursts, or acting aggressively? | 0 0 | 0 | 0 | 0 | 0 |
| Trouble experiencing positive feelings (for example, being unable to feel happiness or have loving feelings for people close to you)? Irritable behavior, angry outbursts, or acting aggressively? Taking too many risks or doing things that could cause you harm? | 0 0 0 | 0 0 0 | 0 0 0 | 0 0 0 | 0 0 0 |
| Trouble experiencing positive feelings (for example, being unable to feel happiness or have loving feelings for people close to you)? Irritable behavior, angry outbursts, or acting aggressively? Taking too many risks or doing things that could cause you harm? Being "superalert" or watchful or on guard? | 0 0 0 0 | 0 0 0 0 | 0 0 0 | 0 0 0 | 0 0 0 |
| Feeling distant or cut off from other people? Trouble experiencing positive feelings (for example, being unable to feel happiness or have loving feelings for people close to you)? Irritable behavior, angry outbursts, or acting aggressively? Taking too many risks or doing things that could cause you harm? Being "superalert" or watchful or on guard? Feeling jumpy or easily startled? Having difficulty concentrating? | 0 0 0 0 0 | 0 0 0 0 0 | 0 0 0 0 0 | 0 0 0 0 0 | 0 0 0 0 0 |
| Trouble experiencing positive feelings (for example, being unable to feel happiness or have loving feelings for people close to you)? Irritable behavior, angry outbursts, or acting aggressively? Taking too many risks or doing things that could cause you harm? Being "superalert" or watchful or on guard? Feeling jumpy or easily startled? | 0 0 0 0 0 0 | 0 0 0 0 0 0 | 0 0 0 0 0 0 | 0 0 0 0 0 0 | 0 0 0 0 0 0 |
| Trouble experiencing positive feelings (for example, being unable to feel happiness or have loving feelings for people close to you)? Irritable behavior, angry outbursts, or acting aggressively? Taking too many risks or doing things that could cause you harm? Being "superalert" or watchful or on guard? Feeling jumpy or easily startled? Having difficulty concentrating? | 0 0 0 0 0 0 | 0 0 0 0 0 0 | 0 0 0 0 0 0 | 0 0 0 0 0 0 | 0 0 0 0 0 0 |

| What is your weight (in pounds)? (If pregnant, please use pre-pregnancy weight.) |
|---|
| RQoL (Health Related Quality of Life) |
| Would you say that in general your health is — |
| Excellent |
| ○ Very good |
| ○ Good |
| ○ Fair |
| O Poor |
| On't know/not sure |
| many days during the <b>past 30 days</b> was your physical health <b>not good</b> ? |
| Now thinking about your <b>mental health</b> , which includes stress, depression, and problems with emotions, for how many days during the <b>past 30 days</b> was your mental health <b>not good</b> ? |
| During the <u>past 30 days</u> , for about how many days did <u>poor physical or mental health</u> keep you from doing your usual activities, such as self care, work, or recreation? |

# AD (Autoimmune Disease)

| Has a doctor, nurse, or other health professional ever diagnosed you with an <u>autoimmune</u> <u>disease</u> ? (e.g., rheumatoid arthritis, hashimoto's disease, Sjogren's syndrome, multiple sclerosis, type 1 |
|---|
| diabetes, systemic lupus erythematosus) |
| ○ No |
| Yes, I have been diagnosed with: |

# PHQ-15 (Somatic Symptoms Survey)

| How much have you been bothered by any of the | ne following probl | ems? | |
|---|---|---|---|
| | Not bothered at all | Bothered a little | Bothered a lo |
| Stomach pain | 0 | 0 | 0 |
| Back pain | 0 | 0 | $\circ$ |
| Pain in your arms, legs, or joints (knees, hips, etc.) | 0 | 0 | 0 |
| Menstrual cramps or other problems with your periods [Women only] | 0 | 0 | 0 |
| Headaches | 0 | 0 | 0 |
| Chest pain | 0 | 0 | 0 |
| Dizziness | 0 | 0 | 0 |
| Fainting spells | 0 | 0 | 0 |
| Feeling your heart pound or race | 0 | 0 | 0 |
| Shortness of breath | 0 | 0 | 0 |
| Pain or problems during sexual intercourse | 0 | 0 | $\circ$ |
| Constipation, loose bowels, or diarrhea | 0 | 0 | $\circ$ |
| Nausea, gas, or indigestion | 0 | 0 | 0 |
| Feeling tired or having low energy | 0 | 0 | $\circ$ |
| Trouble sleeping | 0 | 0 | 0 |

# AUDIT (Alcohol)

The following are questions about your alcohol use in the past 12 months.

A downward of the second of th

| | Never | Less than monthly | Monthly | Weekly | Daily or<br>almost<br>daily |
|---|---|---|---|---|---|
| How often do you have four or more drinks on one occasion? | 0 | 0 | 0 | 0 | 0 |
| How often during the last year have you found that you are not able to stop drinking once you have started? | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| How often during the last year have you failed to do what was normally expected from you because of drinking? | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| How often during the last year have you needed a first drink in the morning to get yourself going after a heavy drinking session? | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| How often during the last year have you had a feeling of guilt or remorse after drinking? | 0 | 0 | 0 | $\circ$ | $\circ$ |
| How often during the last year have you been unable to remember what happened the night before because you had been drinking? | 0 | 0 | 0 | $\circ$ | $\circ$ |

| In the past 12 months | | | |
|---|---|---|---|
| | No | Yes, but not in the last year | Yes, during the last year |
| Have you or someone else been injured as a result of your drinking? | 0 | 0 | 0 |
| Has a relative or friend or doctor or health worker been concerned about your | | | |

5 or 6 7 to 9

10 or more

| The following are questions about other s | ubatanaa uaa | | | | | |
|---|---|---|---|---|---|---|
| | ubstance use | | | | | |
| In the <b>past 12 months</b> , how often have y | /ou | | | | | |
| | | Never | Less than monthly | Monthly | Weekly | Daily o<br>almos<br>daily |
| Jsed any tobacco product (for example, cigarettes, ecigarettes, mokeless tobacco)? | cigars, pipes, or | 0 | 0 | 0 | 0 | 0 |
| Jsed marijuana? | | 0 | 0 | 0 | 0 | 0 |
| Used any prescription medications just for the feeling, more than vere not prescribed for you? | prescribed or that | 0 | 0 | 0 | 0 | 0 |
| Used any other drugs including cocaine or crack, heroin, meth, hecstasy/MDMA? | allucinogens, | 0 | 0 | $\circ$ | $\circ$ | 0 |
| (Sleep Disturbance) | | | | | | |
| | Not at all | 1-3 days | | 8-14 days | 15-21 days | 22-31 da |
| In the <b>past month</b> , did you Have trouble falling asleep? | Not at all | 1-3 days | 4-7 days | 8-14 days | 15-21 days | 22-31 da |
| In the <b>past month</b> , did you Have trouble falling asleep? Wake up several times per night? | Not at all | 1-3 days | | 8-14 days | 15-21 days | 22-31 da |
| In the past month, did you Have trouble falling asleep? Vake up several times per night? Have trouble staying asleep (including waking far too early)? | 0 0 | 1-3 days | | 8-14 days | 15-21 days | 22-31 da |
| In the <b>past month</b> , did you Have trouble falling asleep? Vake up several times per night? Have trouble staying asleep (including waking far too early)? Vake up after your usual amount of sleep feeling tired and worn | 0 0 | 1-3 days | | 8-14 days | 15-21 days | 22-31 da |
| In the <b>past month</b> , did you Have trouble falling asleep? Vake up several times per night? Have trouble staying asleep (including waking far too early)? Vake up after your usual amount of sleep feeling tired and worn out? | 0 0 | 1-3 days | | 8-14 days | 15-21 days | 22-31 da |
| In the <b>past month</b> , did you Have trouble falling asleep? Vake up several times per night? Have trouble staying asleep (including waking far too early)? Vake up after your usual amount of sleep feeling tired and worn out? | 0 0 | 1-3 days | | 8-14 days | 15-21 days | 22-31 da |
| In the past month, did you Have trouble falling asleep? Wake up several times per night? Have trouble staying asleep (including waking far too early)? Wake up after your usual amount of sleep feeling tired and worn out? D-7 (Anxiety) | 0 0 | 1-3 days | | 8-14 days | 15-21 days | 22-31 d |

| The state of the s | | | | 8/6/19, |
|---|---|---|---|---|
| Not being able to stop or control worrying. | ( | 0 | 0 | 0 |
| Worrying too much about different things. | ( | 0 | 0 | 0 |
| Trouble relaxing. | ( | 0 | 0 | $\circ$ |
| Being so restless that it is hard to sit still. | ( | 0 | 0 | $\circ$ |
| Becoming easily annoyed or irritable. | ( | 0 | 0 | $\circ$ |
| Feeling afraid as if something awful might happen. | ( | 0 | 0 | 0 |
| Q-8 (Depression) Over the <u>last two weeks</u> , how often have you bee problems? | n bothered | by any of tl | ne following | |
| Indicate how often any of the following problems ha | | | More than half | Nearly every |
| ittle interest or pleasure doing things | Not at all | Several days | the days | day |
| LILIE INTELESI OF DIEASUFE GOING THINGS. | | | | |
| | 0 | $\circ$ | | |
| Feeling down, depressed, or hopeless. | 0 | 0 | 0 | 0 |
| Feeling down, depressed, or hopeless. Trouble falling or staying asleep, or sleeping too much. | 0 0 | 0 | 0 | 0 |
| Feeling down, depressed, or hopeless. Frouble falling or staying asleep, or sleeping too much. Feeling tired or having little energy. | 0 0 0 | 0 0 0 | 0 0 0 | 0 0 0 |
| Feeling down, depressed, or hopeless. Trouble falling or staying asleep, or sleeping too much. Feeling tired or having little energy. Poor appetite or overeating. Feeling bad about yourself - or that you are a failure or have let yourself or | 0 0 0 0 | 0 0 0 0 | 0 0 0 0 | 0 0 0 |
| Feeling down, depressed, or hopeless. Trouble falling or staying asleep, or sleeping too much. Feeling tired or having little energy. Poor appetite or overeating. Feeling bad about yourself - or that you are a failure or have let yourself or your family down. Trouble concentrating on things, such as reading the newspaper or | 000000 | 0 0 0 0 | 0 0 0 0 | 0 0 0 0 |
| Little interest or pleasure doing things. Feeling down, depressed, or hopeless. Trouble falling or staying asleep, or sleeping too much. Feeling tired or having little energy. Poor appetite or overeating. Feeling bad about yourself - or that you are a failure or have let yourself or your family down. Trouble concentrating on things, such as reading the newspaper or watching television. Moving or speaking so slowly that other people could have noticed. Or the opposite - being so fidgety or restless that you have been moving around a lot more than usual. | 000000 | 000000 | 000000 | 000000 |

# IRI (Empathy)

| | Does not describe me well | 2 | 3 | 4 | Does<br>describe<br>me well |
|---|---|---|---|---|---|
| I daydream and fantasize, with some regularity, about things that might happen to me. | 0 | 0 | 0 | 0 | 0 |
| I often have tender, concerned feelings for people less fortunate than me. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| I sometimes find it difficult to see things from the "other person's" point of view. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Sometimes I don't feel very sorry for other people when they are having problems. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| I really get involved with the feelings of the characters in a novel. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| In emergency situations, I feel apprehensive and ill-at-ease. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I am usually objective when I watch a movie or play, and I don't often get completely caught up in it. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| I try to look at everybody's side of a disagreement before I make a decision. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| When I see someone being taken advantage of, I feel kind of protective towards them. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| I sometimes feel helpless when I am in the middle of a very emotional situation. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| I sometimes try to understand my friends better by imagining how things look from their perspective. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Becoming extremely involved in a good book or movie is somewhat rare for me. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| When I see someone get hurt, I tend to remain calm. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Other people's misfortunes do not usually disturb me a great deal. | 0 | $\circ$ | $\circ$ | 0 | 0 |

| For each item, indicate how well it describes you. | | | | | |
|---|---|---|---|---|---|
| | Does not describe me well | 2 | 3 | 4 | Does<br>describe<br>me well |
| If I'm sure I'm right about something, I don't waste much time listening to other people's arguments. | 0 | 0 | 0 | 0 | 0 |
| After seeing a play or movie, I have felt as though I were one of the characters. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Being in a tense emotional situation scares me. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| When I see someone being treated unfairly, I sometimes don't feel very much pity for them. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I am usually pretty effective in dealing with emergencies. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I am often quite touched by things that I see happen. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| I believe that there are two sides to every question and try to look at them both. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| I would describe myself as a pretty soft-hearted person. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| When I watch a good movie, I can very easily put myself in the place of a leading character. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| I tend to lose control during emergencies. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| When I'm upset at someone, I usually try to "put myself in his shoes" for a while. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| When I am reading an interesting story or novel, I imagine how I would feel if the events in the story were happening to me. | 0 | 0 | 0 | 0 | 0 |

| Before criticizing somebody, I try to imagine how I would feel if I were in their place. | 0 | 0 | 0 | | 0 |
|---|---|---|---|---|---|
| SS Adverse Childhood Experiences (ACEs) | | | | | |
| Next are some questions about events that happened <u>during your childlinformation</u> will allow us to better understand problems that may occur ea help others in the future. <u>Trigger warning</u> . This is a sensitive topic and suncomfortable with these questions. Please keep in mind that you can ski do not want to answer. All questions refer to the time period before you w | rly in<br>ome<br>p any | life<br>peop<br>y qu | and<br>ole m<br>estio | ay f<br>n yo | eel<br>u |
| Now, looking back before you were 18 years of age | | | | | |
| | | | No Ye | kne | Don't<br>ow/no<br>sure |
| Did you live with anyone who was depressed, mentally ill, or suicidal? | | ( | 0 0 | ) | 0 |
| Did you live with anyone who was a problem drinker or alcoholic? | | ( | 0 0 | ) | $\circ$ |
| Did you live with anyone who used illegal street drugs or who abused prescription medications? | | ( | 0 0 | ) | $\circ$ |
| Did you live with anyone who served time or was sentenced to serve time in a prison, jail, or other correctional fac | ility? | | 0 0 | | $\bigcirc$ |
| Now, looking back before you were 18 years of age | No | Vos | Don<br>know/r | not | not |
| Now, looking back before you were 18 years of age Were your parents separated or divorced? | No O | Yes | | not | not |
| | No | Yes | know/ | not | not<br>narried |
| Were your parents separated or divorced? | No | Yes | know/ | not<br>e m | Mor |
| Were your parents separated or divorced? Now, looking back before you were 18 years of age | No | Yes | know/r<br>sure | not<br>e m | not<br>narried<br>Mor<br>thai |
| Were your parents separated or divorced? Now, looking back before you were 18 years of age How often did your parents or adults in your home ever slap, hit, kick, punch or beat each other up? How often did a parent or adult in your home ever hit, beat, kick, or physically hurt you in any way? Do not include | 0 | Yes | know/r<br>sure | not<br>e m | not<br>narried<br>Mor<br>that |
| Were your parents separated or divorced? Now, looking back before you were 18 years of age How often did your parents or adults in your home ever slap, hit, kick, punch or beat each other up? How often did a parent or adult in your home ever hit, beat, kick, or physically hurt you in any way? Do not include spanking. | 0 | Yes | know/r<br>sure | not<br>e m | not<br>narried<br>Mor<br>thai |
| Were your parents separated or divorced? | 0 | Yes | know/r<br>sure | not<br>e m | not<br>narried<br>Mor<br>that |
| Were your parents separated or divorced? Now, looking back before you were 18 years of age How often did your parents or adults in your home ever slap, hit, kick, punch or beat each other up? How often did a parent or adult in your home ever hit, beat, kick, or physically hurt you in any way? Do not include spanking. How often did a parent or adult in your home ever swear at you, insult you, or put you down? | 0 | Yes | know/r<br>sure | not<br>e m | not<br>narrie |

## BRS (Resilience)

| Please respond to each item by selecting one | response be | low. | | | |
|---|---|---|---|---|---|
| | Strongly disagree | Disagree | Neutral | Agree | Strongly agree |
| I tend to bounce back quickly after hard times. | 0 | 0 | 0 | 0 | 0 |
| I have a hard time making it through stressful events. | 0 | 0 | 0 | 0 | 0 |
| It does not take me long to recover from a stressful event. | 0 | 0 | 0 | 0 | 0 |
| It is hard for me to snap back when something bad happens. | 0 | 0 | 0 | 0 | 0 |
| I usually come through difficult times with little trouble. | 0 | 0 | 0 | 0 | 0 |
| I tend to take a long time to get over set-backs in my life. | 0 | 0 | 0 | 0 | 0 |

# ECR-RS (Experiences in Close Relationships - Relationship Structures)

Please read each of the following statements and rate the extent to which you believe each statement best describes your feelings about **close relationships in general**.

| | Strongly disagree | 2 | 3 | 4 | 5 | 6 | Strongly<br>agree |
|---|---|---|---|---|---|---|---|
| It helps to turn to people in times of need. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| I usually discuss my problems and concerns with others. | 0 | $\circ$ | $\circ$ | 0 | $\circ$ | $\circ$ | $\circ$ |
| talk things over with people. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| find it easy to depend on others. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | 0 | $\circ$ |
| don't feel comfortable opening up to others. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 | 0 | $\circ$ |
| prefer not to show others how I feel deep down. | 0 | $\circ$ | 0 | 0 | 0 | 0 | $\circ$ |
| often worry that other people do not really care for me. | 0 | $\circ$ | $\circ$ | 0 | 0 | $\circ$ | $\circ$ |
| 'm afraid that other people may abandon me. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | 0 | $\circ$ |
| worry that others won't care about me as much as I care about them. | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

## MAIA (Interoceptive Awareness)

Below you will find a list of statements.

Please indicate how often each statement applies to you generally in daily life:

| | Never | 1 | 2 | 3 | 4 | Always |
|---|---|---|---|---|---|---|
| When I am tense I notice where the tension is located in my body. | 0 | 0 | 0 | 0 | 0 | 0 |
| I notice when I am uncomfortable in my body. | 0 | $\circ$ | 0 | 0 | $\circ$ | 0 |
| I notice where in my body I am comfortable. | 0 | 0 | 0 | $\circ$ | | $\circ$ |
| I notice changes in my breathing, such as whether it slows down or speeds up. | 0 | $\circ$ | $\circ$ | 0 | 0 | 0 |
| I ignore physical tension or discomfort until they become more severe. | 0 | $\circ$ | $\circ$ | 0 | 0 | 0 |
| I distract myself from sensations of discomfort. | 0 | 0 | 0 | 0 | $\circ$ | 0 |
| When I feel pain or discomfort, I try to power through it. | 0 | $\circ$ | $\circ$ | 0 | 0 | 0 |
| I try to ignore pain. | 0 | 0 | 0 | 0 | $\circ$ | $\circ$ |
| I push feelings of discomfort away by focusing on something. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 | 0 |
| When I feel unpleasant body sensations, I occupy myself with something else so I don't have to feel them. | 0 | 0 | 0 | 0 | 0 | 0 |
| When I feel physical pain, I become upset. | 0 | 0 | 0 | 0 | $\circ$ | 0 |
| I start to worry that something is wrong if I feel any discomfort. | 0 | 0 | 0 | 0 | 0 | 0 |

| Below you will find a | a list | of: | statements. |
|-----------------------|--------|-----|-------------|
|-----------------------|--------|-----|-------------|

Please indicate how often each statement applies to you generally in daily life:

| | • • | • | | • | | |
|---|---|---|---|---|---|---|
| | Never | 1 | 2 | 3 | 4 | Always |
| I can notice an unpleasant body sensation without worrying about it. | 0 | 0 | 0 | 0 | 0 | 0 |
| I can stay calm and not worry when I have feelings of discomfort or pain. | 0 | 0 | $\circ$ | $\circ$ | $\circ$ | 0 |
| When I am in discomfort or pain I can't get it out of my mind. | 0 | $\circ$ | 0 | $\circ$ | 0 | $\circ$ |
| I can pay attention to my breath without being distracted by things happening around me. | 0 | 0 | $\circ$ | $\circ$ | 0 | 0 |
| I can maintain awareness of my inner bodily sensations even when there is a lot going on around me. | 0 | 0 | 0 | 0 | 0 | 0 |
| When I am in conversation with someone, I can pay attention to my posture. | 0 | 0 | $\circ$ | $\circ$ | 0 | 0 |
| I can return awareness to my body if I am distracted. | 0 | $\circ$ | 0 | 0 | $\circ$ | |
| I can refocus my attention from thinking to sensing my body. | 0 | 0 | $\circ$ | $\circ$ | 0 | 0 |
| I can maintain awareness of my whole body even when a part of me is in pain or discomfort. | 0 | 0 | $\circ$ | $\circ$ | 0 | 0 |
| I am able to consciously focus on my body as a | 0 | | | | | |

| | | | | | | _ |
|---|---|---|---|---|---|---|
| notice how my body changes when I am angry. | 0 | 0 | 0 | 0 | 0 | 0 |
| hen something is wrong in my life I can feel it in y body. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| notice that my body feels different after a peaceful kperience. | 0 | 0 | 0 | 0 | 0 | 0 |
| Below you will find a list of statem<br>Please indicate how often each st | | lies to you | ganarally | v in doily l | ifo | |
| rease mulcate now often each st | Never | 1 | 2 | 3 | 4 | Always |
| notice that my breathing becomes free and easy nen I feel comfortable. | 0 | 0 | 0 | 0 | 0 | 0 |
| notice how my body changes when I feel happy / yful. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 | 0 |
| 'hen I feel overwhelmed I can find a calm place<br>side. | 0 | 0 | 0 | 0 | 0 | 0 |
| hen I bring awareness to my body I feel a sense calm. | 0 | $\circ$ | $\circ$ | $\circ$ | 0 | 0 |
| can use my breath to reduce tension. | 0 | 0 | 0 | 0 | 0 | 0 |
| /hen I am caught up in thoughts, I can calm my ind by focusing on my body/breathing. | 0 | 0 | $\circ$ | $\circ$ | 0 | 0 |
| isten for information from my body about my motional state. | 0 | 0 | 0 | 0 | 0 | 0 |
| /hen I am upset, I take time to explore how my ody feels. | 0 | 0 | 0 | 0 | 0 | 0 |
| isten to my body to inform me about what to do. | 0 | 0 | 0 | 0 | 0 | 0 |
| am at home in my body. | 0 | 0 | 0 | 0 | 0 | 0 |
| eel my body is a safe place. | 0 | 0 | 0 | 0 | 0 | 0 |
| rust my body sensations. | 0 | 0 | 0 | 0 | 0 | 0 |

true

true

true

true

true

https://montana.ca1.qualtrics.com/Q/EditSection/Blocks/Ajax/GetSurveyPrintPreview

I criticize myself for having irrational or inappropriate emotions.

I perceive my feelings and emotions without having to react to them.

I'm good at finding words to describe my feelings.

When I'm walking, I deliberately notice the sensations of my body moving.

Qualtrics Survey Software

When I do things, my mind wanders off and I'm easily distracted. 0  $\bigcirc$ 0 0 0 When I take a shower or bath, I stay alert to the sensations of water on my body. I can easily put my beliefs, opinions, and expectations into words. I don't pay attention to what I'm doing because I'm daydreaming, worrying, or otherwise distracted. I watch my feelings without getting lost in them. I tell myself I shouldn't be feeling the way I'm feeling. I notice how foods and drinks affect my thoughts, bodily sensations, and emotions. It's hard for me to find the words to describe what I'm thinking. I am easily distracted. Please select 'Very often' for this response.

| Choose the best response that describes your opinion of what | is gene | erally | true for y | ou. | |
|---|---|---|---|---|---|
| | Never<br>or very<br>rarely<br>true | Rarely<br>true | Sometimes true | Often<br>true | Very<br>often or<br>always<br>true |
| I believe some of my thoughts are abnormal or bad and I shouldn't think that way. | 0 | 0 | 0 | 0 | 0 |
| I pay attention to sensations, such as the wind in my hair or sun on my face. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I have trouble thinking of the right words to express how I feel about things. | 0 | $\circ$ | | $\circ$ | $\circ$ |
| I make judgments about whether my thoughts are good or bad. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| I find it difficult to stay focused on what's happening in the present. | 0 | $\circ$ | | $\circ$ | $\circ$ |
| When I have distressing thoughts or images, I "step back" and am aware of the thought or image without getting taken over by it. | 0 | 0 | $\circ$ | 0 | 0 |
| I pay attention to sounds, such as clocks ticking, birds chirping, or cars passing. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| In difficult situations, I can pause without immediately reacting. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| When I have a sensation in my body, it's difficult for me to describe it because I can't find the right words. | 0 | 0 | $\circ$ | 0 | 0 |
| It seems I am "running on automatic" without much awareness of what I'm doing. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| When I have distressing thoughts or images, I feel calm soon after. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| I tell myself that I shouldn't be thinking the way I'm thinking. | 0 | $\circ$ | | $\circ$ | $\circ$ |
| I notice the smells and aromas of things. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |

| Choose the best response that describes your opinion of what i | s gene | erally t | rue for y | ou. | |
|---|---|---|---|---|---|
| | Never<br>or very<br>rarely<br>true | Rarely<br>true | Sometimes true | Often<br>true | Very<br>often or<br>always<br>true |
| Even when I'm feeling terribly upset, I can find a way to put it into words. | 0 | 0 | 0 | 0 | 0 |

Qualtrics Survey Software

| /hen I have distressing thoughts or images, I just notice them and let them go. do jobs or tasks automatically without being aware of what I'm doing. /hen I have distressing thoughts or images, I judge myself as good or bad, depending what let thought/image is about. pay attention to how my emotions affect my thoughts and behavior. | Survey Software | | | | | |
|---|---|---|---|---|---|---|
| hink some of my emotions are bad or inappropriate and I shouldn't feel them. hotics visual elements in art or nature, such as colors, shapes, textures, or patterns of light dishadow. yo natural tendency is to put my experiences into words. then I have distressing thoughts or images, I just notice them and let them go. do jobs or tasks automatically without being aware of what I'm doing. then I have distressing thoughts or images, I judge myself as good or bad, depending what te thoughthings is about. Dought attention to how my emotions affect my thoughts and behavior. Can usually describe how I feel at the moment in considerable detail. Indimyself doing things without paying attention. Disapprove of myself when I have irrational ideas. Trauma Exposure and Training Questions) Overall, how much of your work involves (directly or indirectly) engaging with traumatized ndividuals or traumatic material? A great deal A lot A moderate amount A little None at all How much training have you received on primary or secondary trauma (including topics like vicarious trauma, secondary traumatic stress, burnout, and moral distress)? A great deal A lot | rush through activities without being really attentive to them. | 0 | 0 | 0 | 0 | 0 |
| notice visual elements in art or nature, such as colors, shapes, textures, or patterns of light dishadow. y natural tendency is to put my experiences into words. hen I have distressing thoughts or images, I just notice them and let them go. to jobs or tasks automatically without being aware of what I'm doing. hen I have distressing thoughts or images, I judge myself as good or bad, depending what et houghtlimage is about. by ay attention to how my emotions affect my thoughts and behavior. van usually describe how I feet at the moment in considerable detail. Ind myself doing things without paying attention. disapprove of myself when I have irrational ideas. Trauma Exposure and Training Questions) Diverall, how much of your work involves (directly or indirectly) engaging with traumatized notividuals or traumatic material? A great deal A lot A moderate amount A little None at all How much training have you received on primary or secondary trauma (including topics like ricarious trauma, secondary traumatic stress, burnout, and moral distress)? A great deal A lot | hen I have distressing thoughts or images I am able just to notice them without reacting. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| Individuals or traumatic material? Agreat deal Alta Agreat deal | hink some of my emotions are bad or inappropriate and I shouldn't feel them. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| then I have distressing thoughts or images, I just notice them and let them go. do jobs or tasks automatically without being aware of what I'm doing. then I have distressing thoughts or images, I judge myself as good or bad, depending what e thought/image is about. apa usually describe how I feel at the moment in considerable detail. and usually describe how I feel at the moment in considerable detail. and myself doing things without paying attention. disapprove of myself when I have irrational ideas. Trauma Exposure and Training Questions) Overall, how much of your work involves (directly or indirectly) engaging with traumatized ndividuals or traumatic material? A great deal A lot A moderate amount A little None at all How much training have you received on primary or secondary trauma (including topics like vicarious trauma, secondary traumatic stress, burnout, and moral distress)? A great deal A lot | | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| do jobs or tasks automatically without being aware of what I'm doing. Then I have distressing thoughts or images, I judge myself as good or bad, depending what et thought/image is about. Day attention to how my emotions affect my thoughts and behavior. Can usually describe how I feel at the moment in considerable detail. Can usually des | ly natural tendency is to put my experiences into words. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Trauma Exposure and Training Questions) Overall, how much of your work involves (directly or indirectly) engaging with traumatized ndividuals or traumatic material? A great deal A little None at all How much training have you received on primary or secondary trauma (including topics like vicarious trauma, secondary traumatic stress, burnout, and moral distress)? A great deal A lot | hen I have distressing thoughts or images, I just notice them and let them go. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| thought/image is about. Doay attention to how my emotions affect my thoughts and behavior. Can usually describe how I feel at the moment in considerable detail. Indiding self doing things without paying attention. Cidisapprove of myself when I have irrational ideas. Trauma Exposure and Training Questions) Overall, how much of your work involves (directly or indirectly) engaging with traumatized individuals or traumatic material? A great deal A lot A moderate amount A little None at all How much training have you received on primary or secondary trauma (including topics like vicarious trauma, secondary traumatic stress, burnout, and moral distress)? A great deal A lot | do jobs or tasks automatically without being aware of what I'm doing. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| can usually describe how I feel at the moment in considerable detail. Inding myself doing things without paying attention. Idisapprove of myself when I have irrational ideas. Trauma Exposure and Training Questions) Overall, how much of your work involves (directly or indirectly) engaging with traumatized individuals or traumatic material? A great deal A lot A moderate amount A little None at all How much training have you received on primary or secondary trauma (including topics like vicarious trauma, secondary traumatic stress, burnout, and moral distress)? A great deal A lot | /hen I have distressing thoughts or images, I judge myself as good or bad, depending what le thought/image is about. | 0 | $\circ$ | 0 | $\circ$ | 0 |
| ind myself doing things without paying attention. disapprove of myself when I have irrational ideas. Trauma Exposure and Training Questions) Overall, how much of your work involves (directly or indirectly) engaging with traumatized ndividuals or traumatic material? A great deal A lot A moderate amount A little None at all How much training have you received on primary or secondary trauma (including topics like vicarious trauma, secondary traumatic stress, burnout, and moral distress)? A great deal A lot | pay attention to how my emotions affect my thoughts and behavior. | 0 | $\circ$ | 0 | 0 | $\circ$ |
| Trauma Exposure and Training Questions) Overall, how much of your work involves (directly or indirectly) engaging with traumatized ndividuals or traumatic material? Agreat deal Alot Amoderate amount Alittle None at all How much training have you received on primary or secondary trauma (including topics like vicarious trauma, secondary traumatic stress, burnout, and moral distress)? Agreat deal Alot | can usually describe how I feel at the moment in considerable detail. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| Trauma Exposure and Training Questions) Overall, how much of your work involves (directly or indirectly) engaging with traumatized ndividuals or traumatic material? Agreat deal Alot A moderate amount A little None at all How much training have you received on primary or secondary trauma (including topics like vicarious trauma, secondary traumatic stress, burnout, and moral distress)? Agreat deal Alot | find myself doing things without paying attention. | 0 | $\circ$ | 0 | $\circ$ | $\circ$ |
| Overall, how much of your work involves (directly or indirectly) engaging with traumatized ndividuals or traumatic material? A great deal A lot A moderate amount A little None at all How much training have you received on primary or secondary trauma (including topics like vicarious trauma, secondary traumatic stress, burnout, and moral distress)? A great deal A lot | disapprove of myself when I have irrational ideas. | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| vicarious trauma, secondary traumatic stress, burnout, and moral distress)? Agreat deal Alot | Overall, how much of your work involves (directly or indirectl ndividuals or traumatic material? | y) engag | ing wit | h traum | atized | |
| A little | Overall, how much of your work involves (directly or indirectl ndividuals or traumatic material? A great deal A lot A moderate amount A little | y) engag | ing wit | h traum | atized | |
| None at all | Overall, how much of your work involves (directly or indirectly ndividuals or traumatic material? A great deal A lot A moderate amount A little None at all How much training have you received on primary or secondary carious trauma, secondary traumatic stress, burnout, and not a great deal A lot A moderate amount | ry trauma | a (inclu | iding to | | e |

Altogether, how effective were your trainings on primary or secondary trauma (including topics

| Extremely effect | ive |
|---|---|
| Very effective | |
| Moderately effect | otive |
| Slightly effective | |
| Not effective at a | |
| o you want<br>econdary tra | more training on secondary trauma (including topics like vicarious trauma, aumatic stress, burnout, and moral distress)? |
| Definitely yes | |
| Probably yes | |
| Might or might n | ot |
| Probably not | |
| Definitely not | |
| Feedback) | y factors affecting your answers that we should know about (e.g., a health issue barrier)? |
| Feedback)<br>Are there any<br>or language I | barrier)? |
| Feedback)<br>Are there any<br>or language I | |
| Feedback)<br>Are there any<br>or language I | barrier)? |

| Thank you for participating in our survey. We would like to email you an Amazon.com eGift Card. To do so, we need you to complete the following questions. |
|---|
| Please allow one week for us to email you the eGift Card. Thanks for your patience with us! |
| What is your first name? |
| What is your last name? |
| What is your phone number (e.g., XXX-XXX-XXXX)? |
| What is your email address? (This is where we will send your e-gift card.) |
| Please verify your email address. |

Official Title: Somatic Mindfulness Training for a Healthy Workforce: Student Pilot Sample

NCT Number: NCT04122534

Document Date: 08/08/2019

## STATISTICAL ANALYSIS PLAN

For each outcome measure (i.e., STSS, PCL-5), most analyses will simply involve calculating descriptive statistics for each wave of data collection. We are pilot testing materials using a small sample and findings will help inform future statistical designs and power needs.